CLINICAL TRIAL: NCT01211652
Title: Gastroprotective Agent Utilization and Compliance in Elderly Patients Taking Non-steroidal Anti-inflammatory Drug (NSAID) in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PFR-DUM-2010/1
Record Dates: First submitted 2010-09-20; First posted 2010-09-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Compliance; France; Self-administered questionnaire to patients
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to assess in general population NSAID and gastroprotective agent utilization and compliance in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* French people > 65 years old, part of Kantar Health Access Santé panel

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 8186 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
NSAID Treatment Compliance | At the end of month 1
Gastroprotective agent compliance (Girerd Questionnaire) | At the end of month 1

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jean-Francois Bretagne, Study Chair — Service gastro-enterologie et hepatologie CHRU Pontchaillou 35033 RENNES cedex France; Pr Gerard Thiefin, Study Chair — Service Hepato-Gastroenterologie CHU Reims 51092 REIMS cedex France; Mrs Genevieve BONNELYE, Principal Investigator — KantarHealth - France138, avenue Marx Dormoy 92120 Montrouge cedex
Locations (3509):
- France (3509):
  - Research Site, Abancourt
  - Research Site, Ablain-Saint-Nazaire
  - Research Site, Ablis
  - Research Site, Ablon-sur-Seine
  - Research Site, Abscon
  - Research Site, Achery
  - Research Site, Achères
  - Research Site, Achicourt
  - Research Site, Achiet-le-Grand
  - Research Site, Adelans-et-le-val-de-bitha
  - Research Site, Adissan
  - Research Site, Agde
  - Research Site, Agen
  - Research Site, Agneaux
  - Research Site, Aiffres
  - Research Site, Aiglun
  - Research Site, Aigrefeuille-sur-Maine
  - Research Site, Aigues-Vives
  - Research Site, Aillevillers-et-Lyaumont
  - Research Site, Ailly-sur-Somme
  - Research Site, Aimargues
  - Research Site, Aime
  - Research Site, Aisey-sur-Seine
  - Research Site, Aix
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Aix-Noulette
  - Research Site, Aixe-sur-Vienne
  - Research Site, Aizier
  - Research Site, Aïssey
  - Research Site, Ajaccio
  - Research Site, Albert
  - Research Site, Albertville
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Alénya
  - Research Site, Alfortville
  - Research Site, Alignan-du-Vent
  - Research Site, Allauch
  - Research Site, Allemans
  - Research Site, Allenjoie
  - Research Site, Alligny-Cosne
  - Research Site, Allonnes
  - Research Site, Alloue
  - Research Site, Almenêches
  - Research Site, Alvimare
  - Research Site, Alzonne
  - Research Site, Amance
  - Research Site, Amancy
  - Research Site, Amanvillers
  - Research Site, Ambazac
  - Research Site, Ambert
  - Research Site, Ambès
  - Research Site, Ambérieu-en-Bugey
  - Research Site, Ambleteuse
  - Research Site, Ambly-sur-Meuse
  - Research Site, Amboise
  - Research Site, Ambrumesnil
  - Research Site, Amfreville-la-Campagne
  - Research Site, Amfreville-les-Champs
  - Research Site, Amiens
  - Research Site, Amilly
  - Research Site, Ancelle
  - Research Site, Ancenis
  - Research Site, Ancerville
  - Research Site, Ancinnes
  - Research Site, Andard
  - Research Site, Andernos-les-Bains
  - Research Site, Andrésy
  - Research Site, Anduze
  - Research Site, Anet
  - Research Site, Anères
  - Research Site, Angers
  - Research Site, Angeville
  - Research Site, Angey
  - Research Site, Angicourt
  - Research Site, Anglars
  - Research Site, Angles
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Angoulins
  - Research Site, Aniche
  - Research Site, Anjouin
  - Research Site, Annecy
  - Research Site, Annecy-le-Vieux
  - Research Site, Annemasse
  - Research Site, Anneville-sur-Mer
  - Research Site, Annoeullin
  - Research Site, Annonay
  - Research Site, Anse
  - Research Site, Anstaing
  - Research Site, Antheny
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Antugnac
  - Research Site, Anzin
  - Research Site, Aouste-sur-Sye
  - Research Site, Appoigny
  - Research Site, Apremont
  - Research Site, Apt
  - Research Site, Aranc
  - Research Site, Arbonne
  - Research Site, Arbonne-la-Forêt
  - Research Site, Arc-lès-Gray
  - Research Site, Arcenant
  - Research Site, Archettes
  - Research Site, Arcueil
  - Research Site, Arçais
  - Research Site, Ardentes
  - Research Site, Aregno
  - Research Site, Arfeuilles
  - Research Site, Argeles
  - Research Site, Argent-sur-Sauldre
  - Research Site, Argentan
  - Research Site, Argentat
  - Research Site, Argenteuil
  - Research Site, Argentré
  - Research Site, Argonay
  - Research Site, Arles
  - Research Site, Arleux
  - Research Site, Armentières
  - Research Site, Arnage
  - Research Site, Arnèke
  - Research Site, Arnouville
  - Research Site, Arpaillargues-et-Aureillac
  - Research Site, Arpajon
  - Research Site, Arques
  - Research Site, Arquian
  - Research Site, Arrancy-sur-Crusnes
  - Research Site, Arras
  - Research Site, Arrènes
  - Research Site, Ars-Laquenexy
  - Research Site, Ars-sur-Moselle
  - Research Site, Arsac
  - Research Site, Arsac-en-Velay
  - Research Site, Artannes-sur-Thouet
  - Research Site, Arthon-en-Retz
  - Research Site, Asasp-Arros
  - Research Site, Ascain
  - Research Site, Asnan
  - Research Site, Asnières-sur-Nouère
  - Research Site, Asnières-sur-Oise
  - Research Site, Asnières-sur-Seine
  - Research Site, Assais-les-Jumeaux
  - Research Site, Astaffort
  - Research Site, Astugue
  - Research Site, Athis-Mons
  - Research Site, Aubagne
  - Research Site, Aubais
  - Research Site, Aubergenville
  - Research Site, Aubervilliers
  - Research Site, Aubevoye
  - Research Site, Aubière
  - Research Site, Aubigné
  - Research Site, Aubigny-sur-Nère
  - Research Site, Aubord
  - Research Site, Auboué
  - Research Site, Aucamville
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Audincourt
  - Research Site, Aulnat
  - Research Site, Aulnay-la-Rivière
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aulnoy
  - Research Site, Aulnoy-lez-Valenciennes
  - Research Site, Aulnoye-Aymeries
  - Research Site, Aumâtre
  - Research Site, Aumetz
  - Research Site, Aumont-Aubrac
  - Research Site, Auray
  - Research Site, Aurec-sur-Loire
  - Research Site, Aureilhan
  - Research Site, Auribeau-sur-Siagne
  - Research Site, Aurillac
  - Research Site, Aussac-Vadalle
  - Research Site, Aussillon
  - Research Site, Auterive
  - Research Site, Authon-Ébéon
  - Research Site, Autignac
  - Research Site, Autun
  - Research Site, Auvers-sur-Oise
  - Research Site, Auxerre
  - Research Site, Auxonne
  - Research Site, Auzainvilliers
  - Research Site, Auzances
  - Research Site, Avanton
  - Research Site, Avelin
  - Research Site, Avermes
  - Research Site, Avesnes-Chaussoy
  - Research Site, Avesnes-le-Comte
  - Research Site, Avesnes-sur-Helpe
  - Research Site, Avignon
  - Research Site, Avion
  - Research Site, Avoine
  - Research Site, Avon
  - Research Site, Ayat-sur-Sioule
  - Research Site, Aytré
  - Research Site, Azay-le-Rideau
  - Research Site, Azelot
  - Research Site, Azereix
  - Research Site, Badonviller
  - Research Site, Bages
  - Research Site, Bagneux
  - Research Site, Bagnolet
  - Research Site, Bagnols-en-Forêt
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baigts-de-Béarn
  - Research Site, Baillet-en-France
  - Research Site, Bailleul
  - Research Site, Bailleul-Sir-Berthoult
  - Research Site, Bailly-Romainvilliers
  - Research Site, Baisieux
  - Research Site, Ballan-Miré
  - Research Site, Ballons
  - Research Site, Balma
  - Research Site, Banassac
  - Research Site, Bangor
  - Research Site, Bar-le-Duc
  - Research Site, Bar-sur-Aube
  - Research Site, Bar-sur-Seine
  - Research Site, Barbentane
  - Research Site, Barberaz
  - Research Site, Barberey-Saint-Sulpice
  - Research Site, Bardenac
  - Research Site, Bardouville
  - Research Site, Barjac
  - Research Site, Barlin
  - Research Site, Barneville-Carteret
  - Research Site, Barr
  - Research Site, Bassens
  - Research Site, Bastia
  - Research Site, Batilly
  - Research Site, Baudoncourt
  - Research Site, Baudreix
  - Research Site, Baule
  - Research Site, Bauné
  - Research Site, Bauvin
  - Research Site, Bayeux
  - Research Site, Bayon
  - Research Site, Bayonne
  - Research Site, Bazancourt
  - Research Site, Bazoches-lès-Bray
  - Research Site, Bazoilles-sur-Meuse
  - Research Site, Beaucaire
  - Research Site, Beaucamps-le-Vieux
  - Research Site, Beauchamps
  - Research Site, Beaufay
  - Research Site, Beaufort
  - Research Site, Beaufort-sur-Gervanne
  - Research Site, Beaugency
  - Research Site, Beaulieu
  - Research Site, Beaulieu-sur-Loire
  - Research Site, Beaulieu-sur-Mer
  - Research Site, Beaulon
  - Research Site, Beaumes-de-Venise
  - Research Site, Beaumé
  - Research Site, Beaumont-du-Ventoux
  - Research Site, Beaumont-sur-Dême
  - Research Site, Beaune
  - Research Site, Beaurains
  - Research Site, Beausoleil
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Beauvallon
  - Research Site, Beauvène
  - Research Site, Beauvoisin
  - Research Site, Behonne
  - Research Site, Belfort
  - Research Site, Belfort-du-Quercy
  - Research Site, Bellac
  - Research Site, Bellaing
  - Research Site, Bellegarde
  - Research Site, Bellegarde-en-Marche
  - Research Site, Bellerive-sur-Allier
  - Research Site, Belleu
  - Research Site, Belleville
  - Research Site, Belley
  - Research Site, Bellême
  - Research Site, Belligné
  - Research Site, Belloy-en-France
  - Research Site, Belrupt
  - Research Site, Bendejun
  - Research Site, Benest
  - Research Site, Benet
  - Research Site, Benfeld
  - Research Site, Benon
  - Research Site, Berck
  - Research Site, Bergueneuse
  - Research Site, Berlaimont
  - Research Site, Bernaville
  - Research Site, Bernay
  - Research Site, Bernières-sur-Mer
  - Research Site, Bernin
  - Research Site, Bernis
  - Research Site, Bernos-Beaulac
  - Research Site, Berre-l'Étang
  - Research Site, Bersée
  - Research Site, Bertangles
  - Research Site, Berthegon
  - Research Site, Berthenay
  - Research Site, Bertoncourt
  - Research Site, Besançon
  - Research Site, Besneville
  - Research Site, Bessancourt
  - Research Site, Bethoncourt
  - Research Site, Bettancourt-la-Ferrée
  - Research Site, Bettant
  - Research Site, Betton
  - Research Site, Beuvry
  - Research Site, Bey
  - Research Site, Beynes
  - Research Site, Beynost
  - Research Site, Bezange-la-Grande
  - Research Site, Bezons
  - Research Site, Bègles
  - Research Site, Bécon-les-Granits
  - Research Site, Bédarieux
  - Research Site, Bédoin
  - Research Site, Bégadan
  - Research Site, Bégard
  - Research Site, Bénaménil
  - Research Site, Bénesse-Maremne
  - Research Site, Béruges
  - Research Site, Bétheniville
  - Research Site, Bétheny
  - Research Site, Béthune
  - Research Site, Bézenet
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Bias
  - Research Site, Bidart
  - Research Site, Bidos
  - Research Site, Bienvillers-au-Bois
  - Research Site, Bièvres
  - Research Site, Biguglia
  - Research Site, Bihorel
  - Research Site, Billère
  - Research Site, Billé
  - Research Site, Billom
  - Research Site, Billy-sur-Aisne
  - Research Site, Bioussac
  - Research Site, Birac
  - Research Site, Biscarrosse
  - Research Site, Bischheim
  - Research Site, Biziat
  - Research Site, Blagnac
  - Research Site, Blain
  - Research Site, Blainville-sur-l'Eau
  - Research Site, Blanchefosse-et-Bay
  - Research Site, Blanquefort
  - Research Site, Blanzac-lès-Matha
  - Research Site, Blanzy-lès-Fismes
  - Research Site, Blasimon
  - Research Site, Blaye
  - Research Site, Blèves
  - Research Site, Blois
  - Research Site, Blotzheim
  - Research Site, Bobigny
  - Research Site, Bohars
  - Research Site, Bois-Colombes
  - Research Site, Bois-de-Céné
  - Research Site, Bois-Guillaume
  - Research Site, Boisredon
  - Research Site, Boissise-la-Bertrand
  - Research Site, Boissise-le-Roi
  - Research Site, Boissy-Saint-Léger
  - Research Site, Bolbec
  - Research Site, Bollène
  - Research Site, Bollwiller
  - Research Site, Bompas
  - Research Site, Bon-Encontre
  - Research Site, Boncé
  - Research Site, Bonchamp-lès-Laval
  - Research Site, Bondoufle
  - Research Site, Bondues
  - Research Site, Bondy
  - Research Site, Bonnard
  - Research Site, Bonnat
  - Research Site, Bonne
  - Research Site, Bonnetan
  - Research Site, Bonneuil-les-Eaux
  - Research Site, Bonneuil-sur-Marne
  - Research Site, Bonneval
  - Research Site, Bonnétable
  - Research Site, Bonsecours
  - Research Site, Bonson
  - Research Site, Bordeaux
  - Research Site, Bordères-sur-l'Échez
  - Research Site, Bosjean
  - Research Site, Bouaye
  - Research Site, Bouc-Bel-Air
  - Research Site, Bouchain
  - Research Site, Boué
  - Research Site, Bougé-Chambalud
  - Research Site, Bougival
  - Research Site, Bouguenais
  - Research Site, Bouillac
  - Research Site, Bouillargues
  - Research Site, Bouilly
  - Research Site, Boujailles
  - Research Site, Boulay-Moselle
  - Research Site, Boulazac
  - Research Site, Boulbon
  - Research Site, Bouligny
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourbon-l'Archambault
  - Research Site, Bourbonne-les-Bains
  - Research Site, Bourbriac
  - Research Site, Bourg-de-Visa
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourg-lès-Valence
  - Research Site, Bourg-Saint-Bernard
  - Research Site, Bourges
  - Research Site, Bourgoin
  - Research Site, Bournezeau
  - Research Site, Bousies
  - Research Site, Boussac
  - Research Site, Bousse
  - Research Site, Boutigny-sur-Essonne
  - Research Site, Bouvesse-Quirieu
  - Research Site, Bouxières-aux-Chênes
  - Research Site, Bouxières-aux-Dames
  - Research Site, Bouy-sur-Orvin
  - Research Site, Bouzillé
  - Research Site, Boves
  - Research Site, Brabant-le-Roi
  - Research Site, Bracieux
  - Research Site, Brainville
  - Research Site, Branoux-les-Taillades
  - Research Site, Brasparts
  - Research Site, Bray-Dunes
  - Research Site, Brech
  - Research Site, Brem-sur-Mer
  - Research Site, Bresles
  - Research Site, Bressuire
  - Research Site, Brest
  - Research Site, Bretenoux
  - Research Site, Bretignolles-sur-Mer
  - Research Site, Bretoncelles
  - Research Site, Brette-les-Pins
  - Research Site, Breuil-la-Réorte
  - Research Site, Breuil-Magné
  - Research Site, Breuillet
  - Research Site, Breux-Jouy
  - Research Site, Brevilliers
  - Research Site, Bréançon
  - Research Site, Bréauté
  - Research Site, Bréhal
  - Research Site, Brétigny-sur-Orge
  - Research Site, Bréval
  - Research Site, Bréviandes
  - Research Site, Briançon
  - Research Site, Brie
  - Research Site, Brie-Comte-Robert
  - Research Site, Briennon
  - Research Site, Brignoles
  - Research Site, Briis-sous-Forges
  - Research Site, Brin-sur-Seille
  - Research Site, Brindas
  - Research Site, Brionne
  - Research Site, Briouze
  - Research Site, Brison-Saint-Innocent
  - Research Site, Brissac
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bron
  - Research Site, Broquiès
  - Research Site, Broussey-Raulecourt
  - Research Site, Bruailles
  - Research Site, Bruay-la-Buissière
  - Research Site, Bruay-sur-l'Escaut
  - Research Site, Bruges
  - Research Site, Bruguières
  - Research Site, Brumath
  - Research Site, Brunoy
  - Research Site, Brunstatt
  - Research Site, Bruville
  - Research Site, Bruyères-et-Montbérault
  - Research Site, Bruz
  - Research Site, Bry-sur-Marne
  - Research Site, Buc
  - Research Site, Bucy-le-Long
  - Research Site, Buis-les-Baronnies
  - Research Site, Buissoncourt
  - Research Site, Bully-les-Mines
  - Research Site, Bures-sur-Yvette
  - Research Site, Burlats
  - Research Site, Bussac-Forêt
  - Research Site, Bussière-Poitevine
  - Research Site, Bussy
  - Research Site, Bussy-Saint-Martin
  - Research Site, Busy
  - Research Site, Butry-sur-Oise
  - Research Site, Buxières-les-Mines
  - Research Site, Buzançais
  - Research Site, Cabariot
  - Research Site, Cabestany
  - Research Site, Cabourg
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cagnotte
  - Research Site, Cagny
  - Research Site, Cahagnes
  - Research Site, Cahors
  - Research Site, Cahuzac
  - Research Site, Calais
  - Research Site, Calenzana
  - Research Site, Calonges
  - Research Site, Calonne-Ricouart
  - Research Site, Caluire-et-Cuire
  - Research Site, Calvisson
  - Research Site, Camaret-sur-Aigues
  - Research Site, Camaret-sur-Mer
  - Research Site, Cambes
  - Research Site, Cambrai
  - Research Site, Camiers
  - Research Site, Camon
  - Research Site, Campan
  - Research Site, Canaples
  - Research Site, Cancale
  - Research Site, Candillargues
  - Research Site, Canet-en-Roussillon
  - Research Site, Canly
  - Research Site, Cannes
  - Research Site, Cannes-Écluse
  - Research Site, Canteleu
  - Research Site, Capbreton
  - Research Site, Capestang
  - Research Site, Cappelle-la-Grande
  - Research Site, Carbon-Blanc
  - Research Site, Carbonne
  - Research Site, Carcassonne
  - Research Site, Carhaix-Plouguer
  - Research Site, Carignan
  - Research Site, Carling
  - Research Site, Carmaux
  - Research Site, Carnoux-en-Provence
  - Research Site, Carolles
  - Research Site, Caromb
  - Research Site, Carpentras
  - Research Site, Carquefou
  - Research Site, Carqueiranne
  - Research Site, Carrières-sous-Poissy
  - Research Site, Carrières-sur-Seine
  - Research Site, Carros
  - Research Site, Carvin
  - Research Site, Cassagnoles
  - Research Site, Cassel
  - Research Site, Cassis
  - Research Site, Casson
  - Research Site, Castanet-Tolosan
  - Research Site, Castellare-di-Casinca
  - Research Site, Castelnau-de-Lévis
  - Research Site, Castelnau-le-Lez
  - Research Site, Castelnau-Magnoac
  - Research Site, Castelnau-Montratier
  - Research Site, Castelnaudary
  - Research Site, Castet
  - Research Site, Castillon-la-Bataille
  - Research Site, Castres
  - Research Site, Castries
  - Research Site, Caudebec-en-Caux
  - Research Site, Caudry
  - Research Site, Caumont-sur-Durance
  - Research Site, Caussens
  - Research Site, Caux
  - Research Site, Cavaillon
  - Research Site, Cavalaire-sur-Mer
  - Research Site, Caylus
  - Research Site, Cayrac
  - Research Site, Cazaubon
  - Research Site, Cazères-sur-l'Adour
  - Research Site, Cazilhac
  - Research Site, Ceintrey
  - Research Site, Cellettes
  - Research Site, Censeau
  - Research Site, Cercoux
  - Research Site, Cergy
  - Research Site, Cervera de la Marenda
  - Research Site, Cesseville
  - Research Site, Cesson-Sévigné
  - Research Site, Cestas
  - Research Site, Ceton
  - Research Site, Cénac
  - Research Site, Chabanais
  - Research Site, Chahaignes
  - Research Site, Chailles
  - Research Site, Chalamont
  - Research Site, Chalautre-la-Grande
  - Research Site, Chaleins
  - Research Site, Chalindrey
  - Research Site, Challans
  - Research Site, Challerange
  - Research Site, Challes-les-Eaux
  - Research Site, Chalon-sur-Saône
  - Research Site, Chalonnes-sur-Loire
  - Research Site, Chamalières
  - Research Site, Chamaret
  - Research Site, Chambéry
  - Research Site, Chambon
  - Research Site, Chambon-sur-Voueize
  - Research Site, Chambourcy
  - Research Site, Chambray-lès-Tours
  - Research Site, Chambrey
  - Research Site, Chamonix
  - Research Site, Chamouillac
  - Research Site, Champagné
  - Research Site, Champagné-les-Marais
  - Research Site, Champcevinel
  - Research Site, Champenoux
  - Research Site, Champforgeuil
  - Research Site, Champier
  - Research Site, Champignelles
  - Research Site, Champigny-sur-Marne
  - Research Site, Champigny-sur-Veude
  - Research Site, Champniers
  - Research Site, Champoly
  - Research Site, Champs-sur-Marne
  - Research Site, Changé
  - Research Site, Chaniers
  - Research Site, Chantecoq
  - Research Site, Chanteloup
  - Research Site, Chanteloup-en-Brie
  - Research Site, Chantepie
  - Research Site, Chantérac
  - Research Site, Chantilly
  - Research Site, Chantonnay
  - Research Site, Chantraine
  - Research Site, Chaource
  - Research Site, Chaponnay
  - Research Site, Chaponost
  - Research Site, Charavines
  - Research Site, Charbonnières-les-Bains
  - Research Site, Chard
  - Research Site, Charentay
  - Research Site, Charentilly
  - Research Site, Charenton-du-Cher
  - Research Site, Charenton-le-Pont
  - Research Site, Charentonnay
  - Research Site, Charleval
  - Research Site, Charleville-Mézières
  - Research Site, Charly
  - Research Site, Charly-Oradour
  - Research Site, Charmes
  - Research Site, Charnay-lès-Mâcon
  - Research Site, Charolles
  - Research Site, Charquemont
  - Research Site, Chartres
  - Research Site, Chasnans
  - Research Site, Chasselay
  - Research Site, Chassors
  - Research Site, Chatou
  - Research Site, Chatuzange-le-Goubet
  - Research Site, Chauffailles
  - Research Site, Chaumes-en-Brie
  - Research Site, Chaumont
  - Research Site, Chaumont-sur-Loire
  - Research Site, Chauny
  - Research Site, Chauvigny
  - Research Site, Chavagnes-en-Paillers
  - Research Site, Chavanoz
  - Research Site, Chaville
  - Research Site, Châlette-sur-Loing
  - Research Site, Châlons-du-Maine
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-Arnoux-Saint-Auban
  - Research Site, Château-d'Olonne
  - Research Site, Château-Gontier
  - Research Site, Château-la-Vallière
  - Research Site, Château-Landon
  - Research Site, Château-Salins
  - Research Site, Château-Thierry
  - Research Site, Châteaubourg
  - Research Site, Châteaubriant
  - Research Site, Châteaudouble
  - Research Site, Châteaudun
  - Research Site, Châteaulin
  - Research Site, Châteauneuf-de-Bordette
  - Research Site, Châteauneuf-de-Gadagne
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châteauneuf-Grasse
  - Research Site, Châteauneuf-la-Forêt
  - Research Site, Châteauneuf-les-Martigues
  - Research Site, Châteauneuf-sur-Charente
  - Research Site, Châteauneuf-sur-Loire
  - Research Site, Châteauroux
  - Research Site, Châtel-sur-Moselle
  - Research Site, Châtelaillon-Plage
  - Research Site, Châteldon
  - Research Site, Châtellerault
  - Research Site, Châtenay-Malabry
  - Research Site, Châtenois-les-Forges
  - Research Site, Châtenoy-le-Royal
  - Research Site, Châtillon
  - Research Site, Châtillon-sur-Chalaronne
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Châtillon-sur-Seine
  - Research Site, Chelles
  - Research Site, Chemiré-sur-Sarthe
  - Research Site, Chenaud
  - Research Site, Chennevières-sur-Marne
  - Research Site, Chenommet
  - Research Site, Chenonceaux
  - Research Site, Cherbourg
  - Research Site, Cherves-Richemont
  - Research Site, Cheval-Blanc
  - Research Site, Chevennes
  - Research Site, Chevillon
  - Research Site, Chevilly
  - Research Site, Chevreaux
  - Research Site, Chevrier
  - Research Site, Chevry-Cossigny
  - Research Site, Chécy
  - Research Site, Chéméré
  - Research Site, Chéu
  - Research Site, Chézy-en-Orxois
  - Research Site, Chignin
  - Research Site, Chilleurs-aux-Bois
  - Research Site, Chilly
  - Research Site, Chindrieux
  - Research Site, Chinon
  - Research Site, Choisey
  - Research Site, Choisy-le-Roi
  - Research Site, Cholet
  - Research Site, Chomérac
  - Research Site, Chouppes
  - Research Site, Chouzé-sur-Loire
  - Research Site, Chusclan
  - Research Site, Ciboure
  - Research Site, Cissac-Médoc
  - Research Site, Civrieux
  - Research Site, Claix
  - Research Site, Clamart
  - Research Site, Clamerey
  - Research Site, Claveyson
  - Research Site, Claye-Souilly
  - Research Site, Clefs-Val d'Anjou
  - Research Site, Clermont
  - Research Site, Clermont-Ferrand
  - Research Site, Clermont-l'Hérault
  - Research Site, Cleyrac
  - Research Site, Clères
  - Research Site, Clémery
  - Research Site, Cléré-les-Pins
  - Research Site, Cléron
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Clisson
  - Research Site, Cloué
  - Research Site, Codognan
  - Research Site, Cognac
  - Research Site, Cognin
  - Research Site, Cogolin
  - Research Site, Collioure
  - Research Site, Collonges-au-Mont-d'Or
  - Research Site, Colmar
  - Research Site, Colmars
  - Research Site, Colombelles
  - Research Site, Colombes
  - Research Site, Colombey-les-Belles
  - Research Site, Colombier
  - Research Site, Colombières
  - Research Site, Colomby-sur-Thaon
  - Research Site, Colomiers
  - Research Site, Coly
  - Research Site, Combronde
  - Research Site, Comines
  - Research Site, Commelle
  - Research Site, Commentry
  - Research Site, Commercy
  - Research Site, Compiègne
  - Research Site, Concarneau
  - Research Site, Conches-sur-Gondoire
  - Research Site, Conchy-les-Pots
  - Research Site, Concots
  - Research Site, Concressault
  - Research Site, Condat-en-Combraille
  - Research Site, Condat-sur-Vienne
  - Research Site, Condé-sur-Iton
  - Research Site, Condrieu
  - Research Site, Conflans-Sainte-Honorine
  - Research Site, Confolens
  - Research Site, Contamine-sur-Arve
  - Research Site, Contes
  - Research Site, Conteville
  - Research Site, Contigné
  - Research Site, Contrevoz
  - Research Site, Corbenay
  - Research Site, Corbie
  - Research Site, Corcelles
  - Research Site, Corcelles-les-Monts
  - Research Site, Cordes-sur-Ciel
  - Research Site, Corenc
  - Research Site, Corme-Royal
  - Research Site, Cormontreuil
  - Research Site, Cornas
  - Research Site, Corneillan
  - Research Site, Cornillé
  - Research Site, Cornillon
  - Research Site, Coron
  - Research Site, Cosmes
  - Research Site, Cosne-Cours-sur-Loire
  - Research Site, Cossé-le-Vivien
  - Research Site, Coti-Chiavari
  - Research Site, Coublevie
  - Research Site, Couchey
  - Research Site, Coucy
  - Research Site, Coudekerque-Branche
  - Research Site, Coudeville-sur-Mer
  - Research Site, Coudrecieux
  - Research Site, Couëron
  - Research Site, Coulaines
  - Research Site, Coulanges-lès-Nevers
  - Research Site, Coulanges-sur-Yonne
  - Research Site, Coulans-sur-Gée
  - Research Site, Coulogne
  - Research Site, Coulommiers
  - Research Site, Coulonces
  - Research Site, Coulonges-sur-lAutize
  - Research Site, Coulounieix-Chamiers
  - Research Site, Cour-Cheverny
  - Research Site, Courbevoie
  - Research Site, Courcelles-lès-Lens
  - Research Site, Courcouronnes
  - Research Site, Courcôme
  - Research Site, Courçon
  - Research Site, Courlaoux
  - Research Site, Cournon-d'Auvergne
  - Research Site, Cours-la-Ville
  - Research Site, Courteilles
  - Research Site, Courtenay
  - Research Site, Courtomer
  - Research Site, Coussey
  - Research Site, Coutençon
  - Research Site, Coutouvre
  - Research Site, Coutras
  - Research Site, Couture-d'Argenson
  - Research Site, Couzeix
  - Research Site, Coye-la-Forêt
  - Research Site, Crainvilliers
  - Research Site, Cran-Gevrier
  - Research Site, Cranves-Sales
  - Research Site, Craon
  - Research Site, Craponne
  - Research Site, Creil
  - Research Site, Creney-près-Troyes
  - Research Site, Crespin
  - Research Site, Cresseveuille
  - Research Site, Creutzwald
  - Research Site, Creuzier-le-Neuf
  - Research Site, Crevin
  - Research Site, Créon
  - Research Site, Crépy-en-Valois
  - Research Site, Créteil
  - Research Site, Crézancy-en-Sancerre
  - Research Site, Criel-sur-Mer
  - Research Site, Criquetot-l'Esneval
  - Research Site, Crissey
  - Research Site, Croissy-sur-Seine
  - Research Site, Croix
  - Research Site, Crolles
  - Research Site, Cros
  - Research Site, Crosne
  - Research Site, Crouy
  - Research Site, Crozon
  - Research Site, Crux-la-Ville
  - Research Site, Cublac
  - Research Site, Cucq
  - Research Site, Cuers
  - Research Site, Cuffies
  - Research Site, Cuffy
  - Research Site, Cuges-les-Pins
  - Research Site, Cugnaux
  - Research Site, Cuincy
  - Research Site, Cusset
  - Research Site, Cussy-les-Forges
  - Research Site, Cutry
  - Research Site, Cysoing
  - Research Site, Dainville
  - Research Site, Damelevières
  - Research Site, Damgan
  - Research Site, Damigny
  - Research Site, Dammarie
  - Research Site, Dammarie-les-Lys
  - Research Site, Dammartin-en-Goële
  - Research Site, Damparis
  - Research Site, Dampierre-sur-Salon
  - Research Site, Damville
  - Research Site, Dangé-Saint-Romain
  - Research Site, Dardilly
  - Research Site, Darnétal
  - Research Site, Dauphin
  - Research Site, Davézieux
  - Research Site, Dax
  - Research Site, Dechy
  - Research Site, Delain
  - Research Site, Delle
  - Research Site, Denain
  - Research Site, Deûlémont
  - Research Site, Décines-Charpieu
  - Research Site, Dégagnac
  - Research Site, Dénezé-sous-Doué
  - Research Site, Déols
  - Research Site, Déville-lès-Rouen
  - Research Site, Didenheim
  - Research Site, Dieffenbach-au-Val
  - Research Site, Dieppe
  - Research Site, Dierre
  - Research Site, Dieue-sur-Meuse
  - Research Site, Dieulefit
  - Research Site, Dieulouard
  - Research Site, Digne-les-Bains
  - Research Site, Digny
  - Research Site, Digoin
  - Research Site, Dijon
  - Research Site, Dinard
  - Research Site, Dinéault
  - Research Site, Dives-sur-Mer
  - Research Site, Divonne-les-Bains
  - Research Site, Dixmont
  - Research Site, Dol-de-Bretagne
  - Research Site, Dole
  - Research Site, Dom-le-Mesnil
  - Research Site, Dombasle-sur-Meurthe
  - Research Site, Dombrot-le-Sec
  - Research Site, Domèvre-en-Haye
  - Research Site, Domfront
  - Research Site, Dommartin-lès-Toul
  - Research Site, Domont
  - Research Site, Dompierre-les-Églises
  - Research Site, Dompierre-sur-Helpe
  - Research Site, Dompierre-sur-Mer
  - Research Site, Donchery
  - Research Site, Doncourt-lès-Conflans
  - Research Site, Donnemarie-Dontilly
  - Research Site, Donnement
  - Research Site, Dordives
  - Research Site, Dornot
  - Research Site, Douai
  - Research Site, Douarnenez
  - Research Site, Douchy
  - Research Site, Doudeville
  - Research Site, Doullens
  - Research Site, Dounoux
  - Research Site, Dourdan
  - Research Site, Douvres-la-Délivrande
  - Research Site, Douvrin
  - Research Site, Douzens
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Draveil
  - Research Site, Dreux
  - Research Site, Droue-sur-Drouette
  - Research Site, Drumettaz
  - Research Site, Duhort-Bachen
  - Research Site, Dunières
  - Research Site, Dunkirk
  - Research Site, Duran
  - Research Site, Durrenbach
  - Research Site, Durrenentzen
  - Research Site, Durtol
  - Research Site, Eaubonne
  - Research Site, Eauze
  - Research Site, Eckbolsheim
  - Research Site, Eclaron-braucourt-sainte-l
  - Research Site, Ecques
  - Research Site, Ectot-l'Auber
  - Research Site, Elbeuf
  - Research Site, Elbeuf-en-Bray
  - Research Site, Embrun
  - Research Site, Enghien-les-Bains
  - Research Site, Ennevelin
  - Research Site, Ennezat
  - Research Site, Entraigues-sur-la-Sorgue
  - Research Site, Entrains-sur-Nohain
  - Research Site, Entrepierres
  - Research Site, Entzheim
  - Research Site, Enveig
  - Research Site, Erbray
  - Research Site, Erbrée
  - Research Site, Ermont
  - Research Site, Ernée
  - Research Site, Erquinghem-Lys
  - Research Site, Erstein
  - Research Site, Escassefort
  - Research Site, Escragnolles
  - Research Site, Esnon
  - Research Site, Espédaillac
  - Research Site, Esquelbecq
  - Research Site, Esquibien
  - Research Site, Essert
  - Research Site, Essertenne-et-Cecey
  - Research Site, Essey-lès-Nancy
  - Research Site, Essômes-sur-Marne
  - Research Site, Estaing
  - Research Site, Estaires
  - Research Site, Esterre
  - Research Site, Estevelles
  - Research Site, Estrablin
  - Research Site, Euilly-et-Lombut
  - Research Site, Excenevex
  - Research Site, Excideuil
  - Research Site, Eybens
  - Research Site, Eynesse
  - Research Site, Eyragues
  - Research Site, Eysines
  - Research Site, Èze
  - Research Site, Échavanne
  - Research Site, Échenoz-la-Méline
  - Research Site, Échillais
  - Research Site, Échirolles
  - Research Site, Éclaires
  - Research Site, Écommoy
  - Research Site, Écouflant
  - Research Site, Écourt-Saint-Quentin
  - Research Site, Écoyeux
  - Research Site, Écrouves
  - Research Site, Écully
  - Research Site, Églisolles
  - Research Site, Égreville
  - Research Site, Égriselles-le-Bocage
  - Research Site, Éguilles
  - Research Site, Élancourt
  - Research Site, Éloie
  - Research Site, Émancé
  - Research Site, Émerchicourt
  - Research Site, Épernay
  - Research Site, Épierre
  - Research Site, Épinal
  - Research Site, Épinay-sous-Sénart
  - Research Site, Épinay-sur-Orge
  - Research Site, Épinay-sur-Seine
  - Research Site, Épineuil-le-Fleuriel
  - Research Site, Épouville
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Éragny
  - Research Site, Étables-sur-Mer
  - Research Site, Étain
  - Research Site, Étampes
  - Research Site, Étaples
  - Research Site, Étouvans
  - Research Site, Étretat
  - Research Site, Étréchy
  - Research Site, Étrépagny
  - Research Site, Étroussat
  - Research Site, Étrœungt
  - Research Site, Évaux-les-Bains
  - Research Site, Évenos
  - Research Site, Évian-les-Bains
  - Research Site, Évreux
  - Research Site, Évron
  - Research Site, Évry
  - Research Site, Ézanville
  - Research Site, Faches-Thumesnil
  - Research Site, Fameck
  - Research Site, Faulquemont
  - Research Site, Fauville-en-Caux
  - Research Site, Faux-la-Montagne
  - Research Site, Faverney
  - Research Site, Faye-dAnjou
  - Research Site, Fayet
  - Research Site, Fayet-le-Château
  - Research Site, Feignies
  - Research Site, Fenain
  - Research Site, Ferney-Voltaire
  - Research Site, Ferrière-la-Grande
  - Research Site, Ferrière-la-Petite
  - Research Site, Ferrières
  - Research Site, Feuquières-en-Vimeu
  - Research Site, Feyzin
  - Research Site, Fère-Champenoise
  - Research Site, Fère-en-Tardenois
  - Research Site, Fécamp
  - Research Site, Féy
  - Research Site, Figeac
  - Research Site, Firminy
  - Research Site, Fitz-James
  - Research Site, Flassans-sur-Issole
  - Research Site, Flavacourt
  - Research Site, Flavigny-sur-Moselle
  - Research Site, Flayosc
  - Research Site, Flers
  - Research Site, Flers-en-Escrebieux
  - Research Site, Fleurance
  - Research Site, Fleurieux-sur-l'Arbresle
  - Research Site, Fleury-les-Aubrais
  - Research Site, Fléville-devant-Nancy
  - Research Site, Flize
  - Research Site, Floirac
  - Research Site, Florentin
  - Research Site, Fluy
  - Research Site, Foix
  - Research Site, Fondettes
  - Research Site, Fonsorbes
  - Research Site, Font-Romeu-Odeillo-Via
  - Research Site, Fontaine
  - Research Site, Fontaine-au-Pire
  - Research Site, Fontaine-Guérin
  - Research Site, Fontaine-la-Soret
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontainebleau
  - Research Site, Fontaines-sur-Saône
  - Research Site, Fontains
  - Research Site, Fontanil-Cornillon
  - Research Site, Fontenay
  - Research Site, Fontenay-aux-Roses
  - Research Site, Fontenay-sous-Bois
  - Research Site, Forbach
  - Research Site, Forcalquier
  - Research Site, Forges-les-Eaux
  - Research Site, Fort-Mardyck
  - Research Site, Fos-sur-Mer
  - Research Site, Fouesnant
  - Research Site, Foug
  - Research Site, Fougerolles
  - Research Site, Fougères
  - Research Site, Foulbec
  - Research Site, Fouqueure
  - Research Site, Fourchambault
  - Research Site, Fourmies
  - Research Site, Fourques
  - Research Site, Fourquevaux
  - Research Site, Fozzano
  - Research Site, Francaltroff
  - Research Site, Franconville
  - Research Site, Freneuse
  - Research Site, Fresnay-sur-Sarthe
  - Research Site, Fresnes
  - Research Site, Fresnes-en-Woëvre
  - Research Site, Fressain
  - Research Site, Fresselines
  - Research Site, Freyming-Merlebach
  - Research Site, Frédéric-Fontaine
  - Research Site, Frégimont
  - Research Site, Fréjus
  - Research Site, Frémonville
  - Research Site, Frévent
  - Research Site, Fricourt
  - Research Site, Froidefontaine
  - Research Site, Frontignan
  - Research Site, Frouard
  - Research Site, Fumay
  - Research Site, Fustérouau
  - Research Site, Fuveau
  - Research Site, Gacé
  - Research Site, Gagny
  - Research Site, Gailhan
  - Research Site, Gaillac
  - Research Site, Galametz
  - Research Site, Gamaches
  - Research Site, Gambsheim
  - Research Site, Ganac
  - Research Site, Gannat
  - Research Site, Gap
  - Research Site, Garches
  - Research Site, Garchizy
  - Research Site, Garchy
  - Research Site, Gardanne
  - Research Site, Gardouch
  - Research Site, Garéoult
  - Research Site, Gargenville
  - Research Site, Garons
  - Research Site, Garrigues
  - Research Site, Garrigues-Sainte-Eulalie
  - Research Site, Gauchy
  - Research Site, Gauriac
  - Research Site, Gazeran
  - Research Site, Geispolsheim
  - Research Site, Genas
  - Research Site, Genay
  - Research Site, Gençay
  - Research Site, Genlis
  - Research Site, Gennes
  - Research Site, Gennevilliers
  - Research Site, Gensac-la-Pallue
  - Research Site, Gentelles
  - Research Site, Gentilly
  - Research Site, Gentioux-Pigerolles
  - Research Site, Germagny
  - Research Site, Germigny-l'Evêque
  - Research Site, Gerstheim
  - Research Site, Géanges
  - Research Site, Gémenos
  - Research Site, Gémigny
  - Research Site, Génébrières
  - Research Site, Générac
  - Research Site, Générest
  - Research Site, Génis
  - Research Site, Gérardmer
  - Research Site, Gétigné
  - Research Site, Ghissignies
  - Research Site, Giberville
  - Research Site, Gien
  - Research Site, Gières
  - Research Site, Gif-sur-Yvette
  - Research Site, Gigean
  - Research Site, Gignac-la-Nerthe
  - Research Site, Gimel-les-Cascades
  - Research Site, Gimont
  - Research Site, Ginasservis
  - Research Site, Girac
  - Research Site, Giromagny
  - Research Site, Gironcourt-sur-Vraine
  - Research Site, Givarlais
  - Research Site, Givet
  - Research Site, Givors
  - Research Site, Givry-en-Argonne
  - Research Site, Glageon
  - Research Site, Glénac
  - Research Site, Glos
  - Research Site, Gometz-la-Ville
  - Research Site, Gommegnies
  - Research Site, Gond-Pontouvre
  - Research Site, Gondecourt
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gonesse
  - Research Site, Gonfreville-lOrcher
  - Research Site, Gornac
  - Research Site, Goudargues
  - Research Site, Gournay-sur-Marne
  - Research Site, Goussaincourt
  - Research Site, Goussainville
  - Research Site, Gouvieux
  - Research Site, Graissessac
  - Research Site, Grand-Charmont
  - Research Site, Grand-Couronne
  - Research Site, Grand-Fort-Philippe
  - Research Site, Grande-Synthe
  - Research Site, Grandpuits-Bailly-Carrois
  - Research Site, Grandrieux
  - Research Site, Grandvillars
  - Research Site, Grans
  - Research Site, Granville
  - Research Site, Grasse
  - Research Site, Gravelines
  - Research Site, Graveson
  - Research Site, Gray
  - Research Site, Grayan
  - Research Site, Grenade
  - Research Site, Grenay
  - Research Site, Grenoble
  - Research Site, Gresswiller
  - Research Site, Gressy
  - Research Site, Greucourt
  - Research Site, Grez-en-Bouère
  - Research Site, Gréasque
  - Research Site, Grézieu-la-Varenne
  - Research Site, Griesheim-sur-Souffel
  - Research Site, Grigny
  - Research Site, Grilly
  - Research Site, Grimaud
  - Research Site, Grisy-Suisnes
  - Research Site, Grosbreuil
  - Research Site, Gruchet-le-Valasse
  - Research Site, Guebwiller
  - Research Site, Guengat
  - Research Site, Guenrouet
  - Research Site, Guerfand
  - Research Site, Guermantes
  - Research Site, Gueutteville-les-Grès
  - Research Site, Guécélard
  - Research Site, Guénange
  - Research Site, Guérande
  - Research Site, Guérard
  - Research Site, Guérigny
  - Research Site, Guichen
  - Research Site, Guignicourt
  - Research Site, Guilherand-Granges
  - Research Site, Guillestre
  - Research Site, Guingamp
  - Research Site, Guinglange
  - Research Site, Guipel
  - Research Site, Guitalens-L'Albarède
  - Research Site, Gujan-Mestras
  - Research Site, Gurunhuel
  - Research Site, Habsheim
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Haillicourt
  - Research Site, Haisnes
  - Research Site, Ham
  - Research Site, Hames-Boucres
  - Research Site, Hangest-sur-Somme
  - Research Site, Hannonville-sous-les-Côtes
  - Research Site, Harcourt
  - Research Site, Hardanges
  - Research Site, Hardecourt-aux-Bois
  - Research Site, Hardinvast
  - Research Site, Harmonville
  - Research Site, Harnes
  - Research Site, Hasnon
  - Research Site, Haubourdin
  - Research Site, Hauterives
  - Research Site, Hauteville-Lompnes
  - Research Site, Havange
  - Research Site, Hayange
  - Research Site, Hazebrouck
  - Research Site, Hede
  - Research Site, Heillecourt
  - Research Site, Heiltz-le-Hutier
  - Research Site, Helfaut
  - Research Site, Hem
  - Research Site, Hendaye
  - Research Site, Hendecourt-lès-Cagnicourt
  - Research Site, Hennecourt
  - Research Site, Herblay-sur-Seine
  - Research Site, Hergnies
  - Research Site, Herm
  - Research Site, Hermanville-sur-Mer
  - Research Site, Herméville-en-Woëvre
  - Research Site, Hestrud
  - Research Site, Hettange-Grande
  - Research Site, Heudebouville
  - Research Site, Heugas
  - Research Site, Hélesmes
  - Research Site, Hénin-Beaumont
  - Research Site, Héric
  - Research Site, Héricourt
  - Research Site, Héricourt-en-Caux
  - Research Site, Hérimoncourt
  - Research Site, Hérouville-Saint-Clair
  - Research Site, Hérouvillette
  - Research Site, Hières-sur-Amby
  - Research Site, Hirson
  - Research Site, Homblières
  - Research Site, Hombourg-Haut
  - Research Site, Horbourg-Wihr
  - Research Site, Hornaing
  - Research Site, Hornoy-le-Bourg
  - Research Site, Houdain
  - Research Site, Houeillès
  - Research Site, Houécourt
  - Research Site, Houilles
  - Research Site, Houplines
  - Research Site, Housseras
  - Research Site, Humbligny
  - Research Site, Hures-la-Parade
  - Research Site, Hyères
  - Research Site, Hœnheim
  - Research Site, Hœrdt
  - Research Site, Ifs
  - Research Site, Igny
  - Research Site, Illiers-Combray
  - Research Site, Illkirch-Graffenstaden
  - Research Site, Illzach
  - Research Site, Indre
  - Research Site, Ingersheim
  - Research Site, Ingré
  - Research Site, Intres
  - Research Site, Isbergues
  - Research Site, Isle
  - Research Site, Issoire
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Itancourt
  - Research Site, Iteuil
  - Research Site, Itteville
  - Research Site, Ivry-sur-Seine
  - Research Site, Izeste
  - Research Site, Île-d'Arz
  - Research Site, Janville
  - Research Site, Janzé
  - Research Site, Jarnac
  - Research Site, Jarny
  - Research Site, Jarrie
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jau-Dignac-et-Loirac
  - Research Site, Jaulnes
  - Research Site, Jaunay-Clan
  - Research Site, Jenlain
  - Research Site, Jeu-les-Bois
  - Research Site, Jeumont
  - Research Site, Joigny
  - Research Site, Joinville-le-Pont
  - Research Site, Jolivet
  - Research Site, Jonage
  - Research Site, Jonquières
  - Research Site, Josse
  - Research Site, Jouarre
  - Research Site, Jouars-Pontchartrain
  - Research Site, Joué-lès-Tours
  - Research Site, Jouy
  - Research Site, Jouy-aux-Arches
  - Research Site, Jouy-en-Josas
  - Research Site, Jouy-le-Potier
  - Research Site, Jouy-sur-Morin
  - Research Site, Joze
  - Research Site, Jugon-les-Lacs
  - Research Site, Juillé
  - Research Site, Jujurieux
  - Research Site, Julianges
  - Research Site, Jumilhac-le-Grand
  - Research Site, Jussy-Champagne
  - Research Site, Juvisy-sur-Orge
  - Research Site, Kerbach
  - Research Site, Kingersheim
  - Research Site, Kirrwiller-bosselshausen
  - Research Site, L'Aigle
  - Research Site, L'Épine
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Herm
  - Research Site, L'Hospitalet-du-Larzac
  - Research Site, L'Hôtellerie
  - Research Site, L'Isle-Adam
  - Research Site, L'Isle-Jourdain
  - Research Site, L'Isle-sur-la-Sorgue
  - Research Site, L'Isle-sur-Serein
  - Research Site, L'Union
  - Research Site, La Barre-de-Monts
  - Research Site, La Bassée
  - Research Site, La Bastide-de-Sérou
  - Research Site, La Baule-Escoublac
  - Research Site, La Baume-Cornillane
  - Research Site, La Bazoche-Gouet
  - Research Site, La Bazoge
  - Research Site, La Bâthie
  - Research Site, La Boisse
  - Research Site, La Bouilladisse
  - Research Site, La Brède
  - Research Site, La Cadière-d'Azur
  - Research Site, La Capelle
  - Research Site, La Celle-Saint-Cloud
  - Research Site, La Celle-Saint-Cyr
  - Research Site, La Chapelaude
  - Research Site, La Chapelle-aux-Naux
  - Research Site, La Chapelle-dArmentières
  - Research Site, La Chapelle-de-Guinchay
  - Research Site, La Chapelle-Gauthier
  - Research Site, La Chapelle-Saint-Étienne
  - Research Site, La Chapelle-Saint-Luc
  - Research Site, La Chapelle-Saint-Mesmin
  - Research Site, La Chapelle-Saint-Sauveur
  - Research Site, La Chapelle-sur-Erdre
  - Research Site, La Chapelle-sur-Loire
  - Research Site, La Chapelle-Villars
  - Research Site, La Charité-sur-Loire
  - Research Site, La Chartre-sur-le-Loir
  - Research Site, La Châtaigneraie
  - Research Site, La Châtre
  - Research Site, La Ciotat
  - Research Site, La Colle-sur-Loup
  - Research Site, La Courtine
  - Research Site, La Côte
  - Research Site, La Crau
  - Research Site, La Crèche
  - Research Site, La Croix-Valmer
  - Research Site, La Fare-les-Oliviers
  - Research Site, La Farlède
  - Research Site, La Faurie
  - Research Site, La Ferté-Bernard
  - Research Site, La Ferté-Macé
  - Research Site, La Ferté-Milon
  - Research Site, La Flèche
  - Research Site, La Forêt-du-Parc
  - Research Site, La Fouillouse
  - Research Site, La Garde
  - Research Site, La Garenne-Colombes
  - Research Site, La Glacerie
  - Research Site, La Grande-Paroisse
  - Research Site, La Guerche-sur-l'Aubois
  - Research Site, La Guérinière
  - Research Site, La Haie-Fouassière
  - Research Site, La Haye-Pesnel
  - Research Site, La Jarrie
  - Research Site, La Laigne
  - Research Site, La Lande-Patry
  - Research Site, La Londe-les-Maures
  - Research Site, La Madeleine
  - Research Site, La Madeleine-de-Nonancourt
  - Research Site, La Magdelaine-sur-Tarn
  - Research Site, La Mailleraye-sur-Seine
  - Research Site, La Mancellière-sur-Vire
  - Research Site, La Membrolle-sur-Choisille
  - Research Site, La Mézière
  - Research Site, La Milesse
  - Research Site, La Motte
  - Research Site, La Motte-d'Aveillans
  - Research Site, La Mulatière
  - Research Site, La Mure
  - Research Site, La Murette
  - Research Site, La Neuve-Lyre
  - Research Site, La Neuville-en-tourne-a-fu
  - Research Site, La Noë-Blanche
  - Research Site, La Pacaudière
  - Research Site, La Péruse
  - Research Site, La Ravoire
  - Research Site, La Réole
  - Research Site, La Riche
  - Research Site, La Rivière-de-Corps
  - Research Site, La Roche-de-Rame
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, La Roque-d'Anthéron
  - Research Site, La Rouge
  - Research Site, La Saulce
  - Research Site, La Saunière
  - Research Site, La Selve
  - Research Site, La Sentinelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Talaudière
  - Research Site, La Teste-de-Buch
  - Research Site, La Tour-du-Pin
  - Research Site, La Trinité
  - Research Site, La Tronche
  - Research Site, La Turballe
  - Research Site, La Valette-du-Var
  - Research Site, La Verdière
  - Research Site, La Verpillière
  - Research Site, La Ville-aux-Dames
  - Research Site, La Ville-Dieu-du-Temple
  - Research Site, La Voulte-sur-Rhône
  - Research Site, La Wantzenau
  - Research Site, Labaroche
  - Research Site, Labastide-Clermont
  - Research Site, Labastide-Esparbairenque
  - Research Site, Labergement-lès-Seurre
  - Research Site, Laborde
  - Research Site, Labourse
  - Research Site, Labruguière
  - Research Site, Labruyère
  - Research Site, Lacanche
  - Research Site, Lacoste
  - Research Site, Lacrouzette
  - Research Site, Ladoix-Serrigny
  - Research Site, Lafrançaise
  - Research Site, Lagarrigue
  - Research Site, Lagnieu
  - Research Site, Lagny-le-Sec
  - Research Site, Lagny-sur-Marne
  - Research Site, Lagord
  - Research Site, LAiguillon-sur-Mer
  - Research Site, Laillé
  - Research Site, Lain
  - Research Site, Laires
  - Research Site, Lalandelle
  - Research Site, Laleu
  - Research Site, Lamalou-les-Bains
  - Research Site, Lamarche-sur-Saône
  - Research Site, Lamastre
  - Research Site, Lamazière-Basse
  - Research Site, Lambersart
  - Research Site, Lambesc
  - Research Site, Lambres-lez-Douai
  - Research Site, Lamotte-Beuvron
  - Research Site, Lamouilly
  - Research Site, Landivisiau
  - Research Site, Landorthe
  - Research Site, Landrévarzec
  - Research Site, Laneuveville-devant-Nancy
  - Research Site, Langeais
  - Research Site, Langey
  - Research Site, Langon
  - Research Site, Langueux
  - Research Site, Lannemezan
  - Research Site, Lannilis
  - Research Site, Lannion
  - Research Site, Lans-en-Vercors
  - Research Site, Lansargues
  - Research Site, Lanuéjouls
  - Research Site, Lanvallay
  - Research Site, Laon
  - Research Site, Lapalisse
  - Research Site, Lapalud
  - Research Site, Laragne-Montéglin
  - Research Site, Larée
  - Research Site, Larmor-Plage
  - Research Site, Laronxe
  - Research Site, Laroque-des-Albères
  - Research Site, Laroque-Timbaut
  - Research Site, Lartigue
  - Research Site, Laruscade
  - Research Site, Lasserre-de-Prouille
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Latresne
  - Research Site, Lattes
  - Research Site, Launaguet
  - Research Site, Laurière
  - Research Site, Lauwin-Planque
  - Research Site, Laval
  - Research Site, Lavaldens
  - Research Site, Lavalette
  - Research Site, Lavaur
  - Research Site, Lavelanet
  - Research Site, Lavernose-Lacasse
  - Research Site, Lavit
  - Research Site, Laxou
  - Research Site, Lazer
  - Research Site, Le Barcarès
  - Research Site, Le Barp
  - Research Site, Le Beausset
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Boullay-les-deux-eglise
  - Research Site, Le Boulou
  - Research Site, Le Bourg-Saint-Léonard
  - Research Site, Le Bourget
  - Research Site, Le Bourget-du-Lac
  - Research Site, Le Bouscat
  - Research Site, Le Bousquet
  - Research Site, Le Bousquet-d'Orb
  - Research Site, Le Breuil
  - Research Site, Le Bugue
  - Research Site, Le Buisson-de-Cadouin
  - Research Site, Le Busseau
  - Research Site, Le Cailar
  - Research Site, Le Cannet
  - Research Site, Le Castéra
  - Research Site, Le Cateau-Cambrésis
  - Research Site, Le Cendre
  - Research Site, Le Chay
  - Research Site, Le Château-d’Oléron
  - Research Site, Le Chesnay
  - Research Site, Le Creusot
  - Research Site, Le Crès
  - Research Site, Le Fossat
  - Research Site, Le Gault-Perche
  - Research Site, Le Gault-Saint-Denis
  - Research Site, Le Genest-Saint-Isle
  - Research Site, Le Gouray
  - Research Site, Le Grand-Abergement
  - Research Site, Le Grand-Bourg
  - Research Site, Le Grand-Quevilly
  - Research Site, Le Gué-de-la-Chaîne
  - Research Site, Le Haillan
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Lardin-Saint-Lazare
  - Research Site, Le Lindois
  - Research Site, Le Luc
  - Research Site, Le Lude
  - Research Site, Le Mans
  - Research Site, Le Mayet-de-Montagne
  - Research Site, Le Mesnil-Durand
  - Research Site, Le Mesnil-en-Thelle
  - Research Site, Le Mesnil-en-Vallée
  - Research Site, Le Mesnil-Esnard
  - Research Site, Le Mesnil-Saint-Denis
  - Research Site, Le Mée-sur-Seine
  - Research Site, Le Mêle-sur-Sarthe
  - Research Site, Le Muy
  - Research Site, Le Neubourg
  - Research Site, Le Palais-sur-Vienne
  - Research Site, Le Pallet
  - Research Site, Le Passage
  - Research Site, Le Perray-en-Yvelines
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Pêchereau
  - Research Site, Le Pian-Médoc
  - Research Site, Le Plessis-Bouchard
  - Research Site, Le Plessis-Robinson
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Poizat
  - Research Site, Le Pontet
  - Research Site, Le Portel
  - Research Site, Le Pradet
  - Research Site, Le Puy-en-Velay
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Revest-les-Eaux
  - Research Site, Le Taillan-Médoc
  - Research Site, Le Temple-sur-Lot
  - Research Site, Le Thou
  - Research Site, Le Torquesne
  - Research Site, Le Touquet-Paris-Plage
  - Research Site, Le Tréport
  - Research Site, Le Val-dAjol
  - Research Site, Le Vernet
  - Research Site, Le Vésinet
  - Research Site, Lecci
  - Research Site, Lecques
  - Research Site, Leers
  - Research Site, Leffrinckoucke
  - Research Site, Leforest
  - Research Site, Lehaucourt
  - Research Site, Leimbach
  - Research Site, Lencloître
  - Research Site, Lenoncourt
  - Research Site, Lens
  - Research Site, Lentilly
  - Research Site, Les Abrets
  - Research Site, Les Angles
  - Research Site, Les Attaques
  - Research Site, Les Brouzils
  - Research Site, Les Cabannes
  - Research Site, Les Clayes-sous-Bois
  - Research Site, Les Croûtes
  - Research Site, Les Eglisottes-et-chalaure
  - Research Site, Les Epesses
  - Research Site, Les Églises-d'Argenteuil
  - Research Site, Les Gets
  - Research Site, Les Grandes-Chapelles
  - Research Site, Les Granges-Gontardes
  - Research Site, Les Herbiers
  - Research Site, Les Hermites
  - Research Site, Les Lilas
  - Research Site, Les Mages
  - Research Site, Les Mathes
  - Research Site, Les Mayons
  - Research Site, Les Mées
  - Research Site, Les Mureaux
  - Research Site, Les Noës-près-Troyes
  - Research Site, Les Ormes
  - Research Site, Les Ormes-sur-Voulzie
  - Research Site, Les Pavillons-sous-Bois
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Pilles
  - Research Site, Les Riceys
  - Research Site, Les Sables-d'Olonne
  - Research Site, Les Ulis
  - Research Site, Les Vans
  - Research Site, Les Villettes
  - Research Site, Lescure
  - Research Site, Lescure-d'Albigeois
  - Research Site, Lesgor
  - Research Site, Lesneven
  - Research Site, Lesquin
  - Research Site, Lestrem
  - Research Site, Leucate
  - Research Site, Leuville-sur-Orge
  - Research Site, Levallois-Perret
  - Research Site, Lezennes
  - Research Site, Lédergues
  - Research Site, Léguevin
  - Research Site, Léguillac-de-lAuche
  - Research Site, Lésigny
  - Research Site, Lézardrieux
  - Research Site, Lherm
  - Research Site, Liart
  - Research Site, Libourne
  - Research Site, Licques
  - Research Site, Liévin
  - Research Site, Liffré
  - Research Site, Lignan-sur-Orb
  - Research Site, Ligny-en-Cambrésis
  - Research Site, Ligueil
  - Research Site, Ligugé
  - Research Site, Lille
  - Research Site, Lillers
  - Research Site, Limalonges
  - Research Site, Limay
  - Research Site, Limeil-Brévannes
  - Research Site, Limoges
  - Research Site, Lingolsheim
  - Research Site, Linxe
  - Research Site, Lisieux
  - Research Site, Lisle-sur-Tarn
  - Research Site, Lisses
  - Research Site, Lissieu
  - Research Site, Listrac-Médoc
  - Research Site, Liverdun
  - Research Site, Livry-Gargan
  - Research Site, Lixy
  - Research Site, Lizières
  - Research Site, Loc-Brévalaire
  - Research Site, Locarn
  - Research Site, Loches
  - Research Site, Locmaria-Plouzané
  - Research Site, Locmariaquer
  - Research Site, Locminé
  - Research Site, Locqueltas
  - Research Site, Locunolé
  - Research Site, Lodève
  - Research Site, Logonna-Daoulas
  - Research Site, Logrian-Florian
  - Research Site, Loisia
  - Research Site, Loison-sous-Lens
  - Research Site, Loisy-sur-Marne
  - Research Site, Lombez
  - Research Site, Lomme
  - Research Site, Lommerange
  - Research Site, Lompret
  - Research Site, Longchamp
  - Research Site, Longeville-lès-Metz
  - Research Site, Longeville-lès-Saint-Avold
  - Research Site, Longjumeau
  - Research Site, Longpont-sur-Orge
  - Research Site, Longueville
  - Research Site, Longueville-sur-Scie
  - Research Site, Longwy
  - Research Site, Lonlay-l'Abbaye
  - Research Site, Lons
  - Research Site, Lons-le-Saunier
  - Research Site, Looberghe
  - Research Site, Loos
  - Research Site, Loos-en-Gohelle
  - Research Site, Looze
  - Research Site, Lorgies
  - Research Site, Lorgues
  - Research Site, Lorient
  - Research Site, Loriol-sur-Drôme
  - Research Site, Lorleau
  - Research Site, Lormaison
  - Research Site, Lormont
  - Research Site, Lorris
  - Research Site, Louannec
  - Research Site, Loubieng
  - Research Site, Loudéac
  - Research Site, Loudun
  - Research Site, Loué
  - Research Site, Louhans
  - Research Site, Lourches
  - Research Site, Lourdes
  - Research Site, Lourmarin
  - Research Site, Louveciennes
  - Research Site, Louvigné-du-Désert
  - Research Site, Louvres
  - Research Site, Louvroil
  - Research Site, Louze
  - Research Site, Lubersac
  - Research Site, Luc
  - Research Site, Lucé
  - Research Site, Lucéram
  - Research Site, Lucheux
  - Research Site, Luçay-le-Mâle
  - Research Site, Luçon
  - Research Site, Ludon-Médoc
  - Research Site, Ludres
  - Research Site, Lue
  - Research Site, Lugon-et-l'Île-du-Carnay
  - Research Site, Luisant
  - Research Site, Lunel
  - Research Site, Lunel-Viel
  - Research Site, Lunéville
  - Research Site, Lure
  - Research Site, Lutterbach
  - Research Site, Lux
  - Research Site, Luxeuil-les-Bains
  - Research Site, Lyon
  - Research Site, Lys-lez-Lannoy
  - Research Site, Mably
  - Research Site, Machecoul
  - Research Site, Maël-Pestivien
  - Research Site, Magnanville
  - Research Site, Magny-le-Désert
  - Research Site, Magny-les-Hameaux
  - Research Site, Magny-Vernois
  - Research Site, Maillé
  - Research Site, Maillot
  - Research Site, Maine-de-Boixe
  - Research Site, Mainvilliers
  - Research Site, Maisdon-sur-Sèvre
  - Research Site, Maisons-Alfort
  - Research Site, Maisons-Laffitte
  - Research Site, Maisonsgoutte
  - Research Site, Maizières-lès-Metz
  - Research Site, Maîche
  - Research Site, Malakoff
  - Research Site, Malaunay
  - Research Site, Malay
  - Research Site, Malemort-sur-Corrèze
  - Research Site, Malesherbes
  - Research Site, Malissard
  - Research Site, Malzéville
  - Research Site, Mamers
  - Research Site, Mamirolle
  - Research Site, Mance
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Mandeure
  - Research Site, Manduel
  - Research Site, Manosque
  - Research Site, Mansle
  - Research Site, Mant
  - Research Site, Mantes-la-Jolie
  - Research Site, Mantes-la-Ville
  - Research Site, Manthelan
  - Research Site, Marac
  - Research Site, Marambat
  - Research Site, Maraussan
  - Research Site, Marbache
  - Research Site, Marcenod
  - Research Site, Marcigny
  - Research Site, Marcillat-en-Combraille
  - Research Site, Marcilly-sur-Vienne
  - Research Site, Marck
  - Research Site, Marcoing
  - Research Site, Marcq-en-Barœul
  - Research Site, Marcy-l'Étoile
  - Research Site, Marçay
  - Research Site, Mareil-sur-Loir
  - Research Site, Marenla
  - Research Site, Marennes
  - Research Site, Mareuil
  - Research Site, Margaux
  - Research Site, Margencel
  - Research Site, Margon
  - Research Site, Marguerittes
  - Research Site, Marignane
  - Research Site, Marigné-Laillé
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marmande
  - Research Site, Marnay
  - Research Site, Marolles-en-Brie
  - Research Site, Maromme
  - Research Site, Marquette-lez-Lille
  - Research Site, Marquillies
  - Research Site, Mars-la-Tour
  - Research Site, Marsac-sur-Don
  - Research Site, Marsais
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseillan
  - Research Site, Marseille
  - Research Site, Marsillargues
  - Research Site, Martel
  - Research Site, Marthod
  - Research Site, Martigues
  - Research Site, Martin-Église
  - Research Site, Martres-sur-Morge
  - Research Site, Marvejols
  - Research Site, Marzan
  - Research Site, Mas-Grenier
  - Research Site, Masny
  - Research Site, Massiac
  - Research Site, Massongy
  - Research Site, Massy
  - Research Site, Matha
  - Research Site, Matzenheim
  - Research Site, Maubeuge
  - Research Site, Mauguio
  - Research Site, Maureillas-las-Illas
  - Research Site, Maurepas
  - Research Site, Mauron
  - Research Site, Mauves
  - Research Site, Mauvezin
  - Research Site, Mauzé-sur-le-Mignon
  - Research Site, Mauzé-Thouarsais
  - Research Site, Maxéville
  - Research Site, Maxou
  - Research Site, Mayenne
  - Research Site, Mazamet
  - Research Site, Mazerulles
  - Research Site, Mâcon
  - Research Site, Meaux
  - Research Site, Megève
  - Research Site, Mehun-sur-Yèvre
  - Research Site, Meillac
  - Research Site, Melesse
  - Research Site, Melun
  - Research Site, Mende
  - Research Site, Mennecy
  - Research Site, Mens
  - Research Site, Mensignac
  - Research Site, Menton
  - Research Site, Mercuès
  - Research Site, Mercy-le-Bas
  - Research Site, Merlas
  - Research Site, Merlimont
  - Research Site, Merten
  - Research Site, Meschers-sur-Gironde
  - Research Site, Mesnil-Clinchamps
  - Research Site, Mesnil-Sellières
  - Research Site, Mesnil-sur-l'Estrée
  - Research Site, Mespuits
  - Research Site, Messac
  - Research Site, Messanges
  - Research Site, Metz
  - Research Site, Meung-sur-Loire
  - Research Site, Meurchin
  - Research Site, Meursac
  - Research Site, Meux
  - Research Site, Meyenheim
  - Research Site, Meylan
  - Research Site, Meymac
  - Research Site, Meynes
  - Research Site, Meyreuil
  - Research Site, Meyrueis
  - Research Site, Meythet
  - Research Site, Meyzieu
  - Research Site, Mécleuves
  - Research Site, Méjannes-le-Clap
  - Research Site, Mélisey
  - Research Site, Ménétréol-sous-Sancerre
  - Research Site, Ménétrol
  - Research Site, Ménigoute
  - Research Site, Mériel
  - Research Site, Mérignac
  - Research Site, Mérindol
  - Research Site, Méry-sur-Oise
  - Research Site, Migennes
  - Research Site, Milhaud
  - Research Site, Millac
  - Research Site, Millas
  - Research Site, Millau
  - Research Site, Mimet
  - Research Site, Mimizan
  - Research Site, Mios
  - Research Site, Mirabel
  - Research Site, Miramas
  - Research Site, Mirande
  - Research Site, Mirandol-Bourgnounac
  - Research Site, Miraumont
  - Research Site, Miré
  - Research Site, Miribel
  - Research Site, Miserey-Salines
  - Research Site, Missé
  - Research Site, Mittois
  - Research Site, Modane
  - Research Site, Moissac
  - Research Site, Moisville
  - Research Site, Molay
  - Research Site, Molières
  - Research Site, Mollégès
  - Research Site, Molompize
  - Research Site, Moloy
  - Research Site, Molsheim
  - Research Site, Monbazillac
  - Research Site, Moncheux
  - Research Site, Monéteau
  - Research Site, Monistrol-sur-Loire
  - Research Site, Monnaie
  - Research Site, Monnières
  - Research Site, Monplaisant
  - Research Site, Mons
  - Research Site, Mons-en-Barœul
  - Research Site, Monsempron
  - Research Site, Monsols
  - Research Site, Mont-de-Marsan
  - Research Site, Mont-le-Vignoble
  - Research Site, Mont-lès-Neufchâteau
  - Research Site, Mont-Louis
  - Research Site, Mont-près-Chambord
  - Research Site, Mont-Saint-Aignan
  - Research Site, Mont-sur-Monnet
  - Research Site, Montady
  - Research Site, Montagny
  - Research Site, Montaigu-de-Quercy
  - Research Site, Montainville
  - Research Site, Montalieu
  - Research Site, Montargis
  - Research Site, Montarnaud
  - Research Site, Montauban
  - Research Site, Montauban-de-Bretagne
  - Research Site, Montauban-de-Luchon
  - Research Site, Montbard
  - Research Site, Montbeton
  - Research Site, Montbéliard
  - Research Site, Montboucher-sur-Jabron
  - Research Site, Montbozon
  - Research Site, Montbrison
  - Research Site, Montceaux-lès-Provins
  - Research Site, Montcuq
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montdidier
  - Research Site, Monteils
  - Research Site, Montenoy
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Montesquieu-Volvestre
  - Research Site, Montesson
  - Research Site, Monteux
  - Research Site, Montégut
  - Research Site, Montélimar
  - Research Site, Montfavet
  - Research Site, Montfermeil
  - Research Site, Montfort-l'Amaury
  - Research Site, Montfort-le-Gesnois
  - Research Site, Montfort-sur-Meu
  - Research Site, Montfort-sur-Risle
  - Research Site, Montgenèvre
  - Research Site, Montgeron
  - Research Site, Monthermé
  - Research Site, Monthou-sur-Cher
  - Research Site, Montignac
  - Research Site, Montignac-Charente
  - Research Site, Montigny-le-Bretonneux
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montigny-lès-Metz
  - Research Site, Montilly-sur-Noireau
  - Research Site, Montireau
  - Research Site, Montlebon
  - Research Site, Montlhéry
  - Research Site, Montlouis-sur-Loire
  - Research Site, Montluçon
  - Research Site, Montluel
  - Research Site, Montmacq
  - Research Site, Montmeyran
  - Research Site, Montmélian
  - Research Site, Montmoreau-Saint-Cybard
  - Research Site, Montmorency
  - Research Site, Montmorillon
  - Research Site, Montmorin
  - Research Site, Montmort
  - Research Site, Montoir-de-Bretagne
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montolieu
  - Research Site, Montpellier
  - Research Site, Montpeyroux
  - Research Site, Montpon-Ménestérol
  - Research Site, Montrabé
  - Research Site, Montreuil
  - Research Site, Montreuil-Bellay
  - Research Site, Montreuil-Juigné
  - Research Site, Montreuil-sur-Lozon
  - Research Site, Montréal
  - Research Site, Montrouge
  - Research Site, Monts
  - Research Site, Montsûrs
  - Research Site, Moon-sur-Elle
  - Research Site, Mordelles
  - Research Site, Moret-sur-Loing
  - Research Site, Moréac
  - Research Site, Morgny-la-Pommeraye
  - Research Site, Morhange
  - Research Site, Morières-lès-Avignon
  - Research Site, Morigny-Champigny
  - Research Site, Morizès
  - Research Site, Morlaix
  - Research Site, Mormoiron
  - Research Site, Mornant
  - Research Site, Morschwiller-le-Bas
  - Research Site, Mortagne-sur-Gironde
  - Research Site, Mortagne-sur-Sèvre
  - Research Site, Morteau
  - Research Site, Mortroux
  - Research Site, Morvillers
  - Research Site, Mostuéjouls
  - Research Site, Mougins
  - Research Site, Mouilleron-le-Captif
  - Research Site, Moulines
  - Research Site, Moulins
  - Research Site, Moulins-Engilbert
  - Research Site, Moulins-lès-Metz
  - Research Site, Mourenx
  - Research Site, Mouroux
  - Research Site, Mousseaux-Neuville
  - Research Site, Moussoulens
  - Research Site, Moustier-en-Fagne
  - Research Site, Mouvaux
  - Research Site, Mouzeuil-Saint-Martin
  - Research Site, Moyenmoutier
  - Research Site, Moyeuvre-Grande
  - Research Site, Muides-sur-Loire
  - Research Site, Mulhouse
  - Research Site, Mulsanne
  - Research Site, Mundolsheim
  - Research Site, Mur-de-Sologne
  - Research Site, Muret
  - Research Site, Murianette
  - Research Site, Murlin
  - Research Site, Murs
  - Research Site, Muzillac
  - Research Site, Myennes
  - Research Site, Nancy
  - Research Site, Nançois-sur-Ornain
  - Research Site, Nandy
  - Research Site, Nangis
  - Research Site, Nangy
  - Research Site, Nans-les-Pins
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nantouillet
  - Research Site, Narbonne
  - Research Site, Naucelle
  - Research Site, Naves
  - Research Site, Nayemont-les-Fosses
  - Research Site, Nazelles-Négron
  - Research Site, Neauphle-le-Château
  - Research Site, Neffiès
  - Research Site, Nersac
  - Research Site, Neufchâtel-en-Bray
  - Research Site, Neufchâtel-Hardelot
  - Research Site, Neufchef
  - Research Site, Neuflize
  - Research Site, Neuilly-en-Sancerre
  - Research Site, Neuilly-en-Thelle
  - Research Site, Neuilly-le-Vendin
  - Research Site, Neuilly-Plaisance
  - Research Site, Neuilly-sur-Marne
  - Research Site, Neuilly-sur-Seine
  - Research Site, Neuvecelle
  - Research Site, Neuves-Maisons
  - Research Site, Neuvicq
  - Research Site, Neuville-aux-Bois
  - Research Site, Neuville-en-Ferrain
  - Research Site, Neuville-lès-Lœuilly
  - Research Site, Neuville-Saint-Amand
  - Research Site, Neuville-Saint-Rémy
  - Research Site, Neuville-Saint-Vaast
  - Research Site, Neuville-sur-Ornain
  - Research Site, Neuvilly
  - Research Site, Neuvy-Deux-Clochers
  - Research Site, Neuvy-sur-Barangeon
  - Research Site, Neuvy-sur-Loire
  - Research Site, Nevers
  - Research Site, Neyron
  - Research Site, Néris-les-Bains
  - Research Site, Nézignan-l'Évêque
  - Research Site, Nice
  - Research Site, Niderhoff
  - Research Site, Niederhausbergen
  - Research Site, Nielles-lès-Ardres
  - Research Site, Nieppe
  - Research Site, Niherne
  - Research Site, Niort
  - Research Site, Nissan-lez-Enserune
  - Research Site, Nitting
  - Research Site, Nîmes
  - Research Site, Noailhac
  - Research Site, Nogent
  - Research Site, Nogent-le-Roi
  - Research Site, Nogent-le-Rotrou
  - Research Site, Nogent-sur-Marne
  - Research Site, Nogent-sur-Oise
  - Research Site, Nogent-sur-Seine
  - Research Site, Nogentel
  - Research Site, Nohic
  - Research Site, Noisy-le-Grand
  - Research Site, Noisy-le-Roi
  - Research Site, Noisy-le-Sec
  - Research Site, Nommay
  - Research Site, Nonville
  - Research Site, Normanville
  - Research Site, Notre-Dame-d'Oé
  - Research Site, Notre-Dame-de-Boisset
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Notre-Dame-des-Landes
  - Research Site, Notre-Dame-des-Millières
  - Research Site, Notre-Dame-du-Pé
  - Research Site, Nouzonville
  - Research Site, Noyal-sous-Bazouges
  - Research Site, Noyelles-sous-Lens
  - Research Site, Noyers-Pont-Maugis
  - Research Site, Noyon
  - Research Site, Nœux-les-Mines
  - Research Site, Oberhausbergen
  - Research Site, Oberhergheim
  - Research Site, Obernai
  - Research Site, Objat
  - Research Site, Occagnes
  - Research Site, Octeville
  - Research Site, Odos
  - Research Site, Offendorf
  - Research Site, Oissel-sur-Seine
  - Research Site, Oletta
  - Research Site, Olivet
  - Research Site, Ollioules
  - Research Site, Olonne-sur-Mer
  - Research Site, Oloron-Sainte-Marie
  - Research Site, Omonville-la-Petite
  - Research Site, Ondefontaine
  - Research Site, Onet-le-Château
  - Research Site, Onzain
  - Research Site, Oraison
  - Research Site, Orange
  - Research Site, Origny-en-Thiérache
  - Research Site, Orleix
  - Research Site, Orléans
  - Research Site, Orléat
  - Research Site, Orliénas
  - Research Site, Orly
  - Research Site, Ormesson-sur-Marne
  - Research Site, Ormoy-la-Rivière
  - Research Site, Ornans
  - Research Site, Oroix
  - Research Site, Orsay
  - Research Site, Orthez
  - Research Site, Ortoncourt
  - Research Site, Orvault
  - Research Site, Osny
  - Research Site, Ossès
  - Research Site, Oudezeele
  - Research Site, Oudon
  - Research Site, Ouilly-le-Vicomte
  - Research Site, Ouistreham
  - Research Site, Oullins
  - Research Site, Ouroux-sur-Saône
  - Research Site, Oye-Plage
  - Research Site, Oyonnax
  - Research Site, Pagny-la-Ville
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paimpol
  - Research Site, Paimpont
  - Research Site, Paizay-le-Chapt
  - Research Site, Palaiseau
  - Research Site, Palaja
  - Research Site, Palaminy
  - Research Site, Palavas-les-Flots
  - Research Site, Palazinges
  - Research Site, Pamiers
  - Research Site, Panazol
  - Research Site, Pannes
  - Research Site, Pantin
  - Research Site, Paray-le-Monial
  - Research Site, Paray-Vieille-Poste
  - Research Site, Parcieux
  - Research Site, Pargny-Filain
  - Research Site, Pargny-sous-Mureau
  - Research Site, Pargny-sur-Saulx
  - Research Site, Paris
  - Research Site, Paris 01 Louvre
  - Research Site, Paris 10eme
  - Research Site, Parmain
  - Research Site, Paron
  - Research Site, Parthenay
  - Research Site, Passavant-la-Rochère
  - Research Site, Passy
  - Research Site, Pau
  - Research Site, Paulin
  - Research Site, Pavilly
  - Research Site, Pechbonnieu
  - Research Site, Peillac
  - Research Site, Pellevoisin
  - Research Site, Peltre
  - Research Site, Pennautier
  - Research Site, Perceneige
  - Research Site, Percy
  - Research Site, Pernes
  - Research Site, Pernes-les-Fontaines
  - Research Site, Perpignan
  - Research Site, Perrecy-les-Forges
  - Research Site, Perreux
  - Research Site, Perriers-en-Beauficel
  - Research Site, Perros-Guirec
  - Research Site, Persac
  - Research Site, Persan
  - Research Site, Pertuis
  - Research Site, Peschadoires
  - Research Site, Pesmes
  - Research Site, Pessac
  - Research Site, Petite-Rosselle
  - Research Site, Peujard
  - Research Site, Peyrelongue-Abos
  - Research Site, Peyriac-de-Mer
  - Research Site, Peyrins
  - Research Site, Peyrouse
  - Research Site, Péaule
  - Research Site, Péchaudier
  - Research Site, Pélissanne
  - Research Site, Pénestin
  - Research Site, Pérenchies
  - Research Site, Péré
  - Research Site, Périgné
  - Research Site, Périgny
  - Research Site, Périgueux
  - Research Site, Pérols
  - Research Site, Péronnas
  - Research Site, Péronne
  - Research Site, Péronne-en-Mélantois
  - Research Site, Pérouges
  - Research Site, Pfastatt
  - Research Site, Piazzole
  - Research Site, Pierrefitte-en-Beauvaisis
  - Research Site, Pierrefitte-sur-Aire
  - Research Site, Pierrefitte-sur-Sauldre
  - Research Site, Pierrefitte-sur-Seine
  - Research Site, Pierrevert
  - Research Site, Pietroso
  - Research Site, Pieusse
  - Research Site, Pignan
  - Research Site, Pignans
  - Research Site, Pineuilh
  - Research Site, Pins-Justaret
  - Research Site, Pipriac
  - Research Site, Pirey
  - Research Site, Pirou
  - Research Site, Pisany
  - Research Site, Pithiviers
  - Research Site, Pitres
  - Research Site, Plabennec
  - Research Site, Plainfaing
  - Research Site, Plaintel
  - Research Site, Plaisance-du-Touch
  - Research Site, Plaisir
  - Research Site, Plan-de-Cuques
  - Research Site, Plancoët
  - Research Site, Plazac
  - Research Site, Pleine-Sève
  - Research Site, Plestan
  - Research Site, Plestin-les-Grèves
  - Research Site, Pleumeur-Gautier
  - Research Site, Pleuven
  - Research Site, Plédran
  - Research Site, Plélan-le-Grand
  - Research Site, Pléneuf-Val-André
  - Research Site, Plénée-Jugon
  - Research Site, Plérin
  - Research Site, Plonéis
  - Research Site, Plouaret
  - Research Site, Ploubazlanec
  - Research Site, Plouër-sur-Rance
  - Research Site, Ploufragan
  - Research Site, Plougastel-Daoulas
  - Research Site, Plougonven
  - Research Site, Plougrescant
  - Research Site, Plouguin
  - Research Site, Plouha
  - Research Site, Plouigneau
  - Research Site, Plouvain
  - Research Site, Plozévet
  - Research Site, Pluvault
  - Research Site, Podensac
  - Research Site, Poggio-di-Nazza
  - Research Site, Poigny-la-Forêt
  - Research Site, Poissy
  - Research Site, Poitiers
  - Research Site, Polincove
  - Research Site, Pomeys
  - Research Site, Pommerit-Jaudy
  - Research Site, Pommiers
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-de-Barret
  - Research Site, Pont-de-Roide
  - Research Site, Pont-du-Casse
  - Research Site, Pont-Farcy
  - Research Site, Pont-Hébert
  - Research Site, Pont-l'Abbé
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pont-l'Évêque
  - Research Site, Pont-Saint-Pierre
  - Research Site, Pont-Sainte-Marie
  - Research Site, Pont-sur-Yonne
  - Research Site, Pontarlier
  - Research Site, Pontault-Combault
  - Research Site, Pontchâteau
  - Research Site, Pontgouin
  - Research Site, Pontivy
  - Research Site, Pontlevoy
  - Research Site, Pontoise
  - Research Site, Pontpoint
  - Research Site, Pontrieux
  - Research Site, Porcelette
  - Research Site, Pordic
  - Research Site, Pornic
  - Research Site, Pornichet
  - Research Site, Port-de-Bouc
  - Research Site, Port-de-Lanne
  - Research Site, Port-en-Bessin-Huppain
  - Research Site, Port-Saint-Louis-du-Rhône
  - Research Site, Port-sur-Saône
  - Research Site, Portes-lès-Valence
  - Research Site, Portet-sur-Garonne
  - Research Site, Ports
  - Research Site, Portvendres
  - Research Site, Potigny
  - Research Site, Pouillon
  - Research Site, Pouilly-les-Nonains
  - Research Site, Pouilly-sur-Loire
  - Research Site, Poulx
  - Research Site, Pouxeux
  - Research Site, Pouylebon
  - Research Site, Prades
  - Research Site, Prayssac
  - Research Site, Pré-en-Pail
  - Research Site, Préchacq-les-Bains
  - Research Site, Précy-sur-Oise
  - Research Site, Prémilhat
  - Research Site, Priaires
  - Research Site, Pringy
  - Research Site, Prinquiau
  - Research Site, Proville
  - Research Site, Provins
  - Research Site, Puget-sur-Argens
  - Research Site, Pugnac
  - Research Site, Puilboreau
  - Research Site, Pujaut
  - Research Site, Pulnoy
  - Research Site, Pulversheim
  - Research Site, Puteaux
  - Research Site, Puttelange-aux-Lacs
  - Research Site, Quarouble
  - Research Site, Quelaines-Saint-Gault
  - Research Site, Quend
  - Research Site, Querrien
  - Research Site, Quesnoy-sur-Deûle
  - Research Site, Questembert
  - Research Site, Quetigny
  - Research Site, Quetteville
  - Research Site, Quiberon
  - Research Site, Quièvrecourt
  - Research Site, Quimper
  - Research Site, Quincy-Voisins
  - Research Site, Quingey
  - Research Site, Quinsac
  - Research Site, Quint-Fonsegrives
  - Research Site, Rabastens-de-Bigorre
  - Research Site, Radinghem-en-Weppes
  - Research Site, Radon
  - Research Site, Rahon
  - Research Site, Rambervillers
  - Research Site, Rambouillet
  - Research Site, Ramonville-Saint-Agne
  - Research Site, Rang-du-Fliers
  - Research Site, Raon-l'Étape
  - Research Site, Razac-sur-lIsle
  - Research Site, Rânes
  - Research Site, Rebais
  - Research Site, Redon
  - Research Site, Regniowez
  - Research Site, Reignac-sur-Indre
  - Research Site, Reillanne
  - Research Site, Reims
  - Research Site, Remiremont
  - Research Site, Remoncourt
  - Research Site, Remouillé
  - Research Site, Renaison
  - Research Site, Rennes
  - Research Site, Renwez
  - Research Site, Retiers
  - Research Site, Rettel
  - Research Site, Revel
  - Research Site, Revelles
  - Research Site, Revin
  - Research Site, Rexpoëde
  - Research Site, Reyrieux
  - Research Site, Rezé
  - Research Site, Réauville
  - Research Site, Réding
  - Research Site, Rémelfang
  - Research Site, Rémilly
  - Research Site, Rians
  - Research Site, Ribaute-les-Tavernes
  - Research Site, Ribeauvillé
  - Research Site, Richardménil
  - Research Site, Richelieu
  - Research Site, Riedisheim
  - Research Site, Riez
  - Research Site, Rigny
  - Research Site, Rigny-le-Ferron
  - Research Site, Rilhac-Rancon
  - Research Site, Rilhac-Xaintrie
  - Research Site, Rillieux-la-Pape
  - Research Site, Riols
  - Research Site, Riom
  - Research Site, Ris-Orangis
  - Research Site, Rives
  - Research Site, Rivesaltes
  - Research Site, Rivière
  - Research Site, Rivières
  - Research Site, Rixheim
  - Research Site, Roanne
  - Research Site, Robion
  - Research Site, Rocbaron
  - Research Site, Roche-la-Molière
  - Research Site, Rochechouart
  - Research Site, Rochefort
  - Research Site, Rochemaure
  - Research Site, Rodilhan
  - Research Site, Rognac
  - Research Site, Rognes
  - Research Site, Rohan
  - Research Site, Roissy-en-Brie
  - Research Site, Roissy-en-France
  - Research Site, Romagnat
  - Research Site, Romainville
  - Research Site, Romans-sur-Isère
  - Research Site, Rombas
  - Research Site, Romilly-sur-Seine
  - Research Site, Romorantin-Lanthenay
  - Research Site, Ronchères
  - Research Site, Ronchin
  - Research Site, Roncq
  - Research Site, Roquebrune-Cap-Martin
  - Research Site, Roquebrune-sur-Argens
  - Research Site, Roquefort-sur-Garonne
  - Research Site, Roquemaure
  - Research Site, Roques
  - Research Site, Roquevaire
  - Research Site, Rosheim
  - Research Site, Rosières
  - Research Site, Rosny-sous-Bois
  - Research Site, Rosny-sur-Seine
  - Research Site, Rosoy-en-Multien
  - Research Site, Rosporden
  - Research Site, Rosult
  - Research Site, Rotalier
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rougemont
  - Research Site, Rougemont-le-Château
  - Research Site, Rougé
  - Research Site, Rouhling
  - Research Site, Rouillac
  - Research Site, Rouillé
  - Research Site, Rouillon
  - Research Site, Roussas
  - Research Site, Routot
  - Research Site, Rouvres-en-Plaine
  - Research Site, Rouvroy
  - Research Site, Royan
  - Research Site, Roz-Landrieux
  - Research Site, Rueil-Malmaison
  - Research Site, Ruelisheim
  - Research Site, Ruelle-sur-Touvre
  - Research Site, Ruffec
  - Research Site, Ruffey-sur-Seille
  - Research Site, Rumilly
  - Research Site, Rungis
  - Research Site, Rupt-sur-Moselle
  - Research Site, Rustenhart
  - Research Site, Sablé-sur-Sarthe
  - Research Site, Sacy
  - Research Site, Sacy-le-Grand
  - Research Site, Saillant
  - Research Site, Saillenard
  - Research Site, Sailly-Labourse
  - Research Site, Sailly-sur-la-Lys
  - Research Site, Sainghin-en-Weppes
  - Research Site, Sainneville
  - Research Site, Sains-en-Gohelle
  - Research Site, Saint Nicolas Les Arras
  - Research Site, Saint-Agathon
  - Research Site, Saint-Agnant
  - Research Site, Saint-Aignan
  - Research Site, Saint-Amand
  - Research Site, Saint-Amand-les-Eaux
  - Research Site, Saint-Amand-Montrond
  - Research Site, Saint-Amant-Tallende
  - Research Site, Saint-Amarin
  - Research Site, Saint-André-de-Cubzac
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-de-Valborgne
  - Research Site, Saint-André-le-Gaz
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Antoine-Cumond
  - Research Site, Saint-Antoine-du-Rocher
  - Research Site, Saint-Antonin-Noble-Val
  - Research Site, Saint-Apollinaire
  - Research Site, Saint-Armel
  - Research Site, Saint-Arnoult
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Astier
  - Research Site, Saint-Auban
  - Research Site, Saint-Aubin-de-Médoc
  - Research Site, Saint-Aubin-du-Cormier
  - Research Site, Saint-Aubin-le-Vertueux
  - Research Site, Saint-Aubin-sur-Gaillon
  - Research Site, Saint-Aubin-sur-Mer
  - Research Site, Saint-Aulaye
  - Research Site, Saint-Avertin
  - Research Site, Saint-Avit
  - Research Site, Saint-Avit-Saint-Nazaire
  - Research Site, Saint-Avold
  - Research Site, Saint-Barthélémy
  - Research Site, Saint-Benoît
  - Research Site, Saint-Benoît-de-Carmaux
  - Research Site, Saint-Benoît-sur-Loire
  - Research Site, Saint-Berthevin
  - Research Site, Saint-Blaise-la-Roche
  - Research Site, Saint-Bohaire
  - Research Site, Saint-Bonnet-de-Mure
  - Research Site, Saint-Briac-sur-Mer
  - Research Site, Saint-Brice-Courcelles
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Bris-des-Bois
  - Research Site, Saint-Calais
  - Research Site, Saint-Caradec
  - Research Site, Saint-Cassien
  - Research Site, Saint-Cernin-de-l'Herm
  - Research Site, Saint-Céré
  - Research Site, Saint-Cézaire-sur-Siagne
  - Research Site, Saint-Chamond
  - Research Site, Saint-Christol-les-Alès
  - Research Site, Saint-Ciers-sur-Bonnieure
  - Research Site, Saint-Clair-de-la-Tour
  - Research Site, Saint-Claud
  - Research Site, Saint-Claude
  - Research Site, Saint-Clément
  - Research Site, Saint-Cloud
  - Research Site, Saint-Contest
  - Research Site, Saint-Cosme-en-Vairais
  - Research Site, Saint-Crespin-sur-Moine
  - Research Site, Saint-Cyprien
  - Research Site, Saint-Cyr-au-Mont-d'Or
  - Research Site, Saint-Cyr-les-Champagnes
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-du-Pin
  - Research Site, Saint-Denis-en-Bugey
  - Research Site, Saint-Denis-en-Val
  - Research Site, Saint-Didier-de-la-Tour
  - Research Site, Saint-didier-sur-chalaronn
  - Research Site, Saint-Dié
  - Research Site, Saint-Dizier
  - Research Site, Saint-Domineuc
  - Research Site, Saint-Donat-sur-l'Herbasse
  - Research Site, Saint-Erblon
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-etienne-les-remiremo
  - Research Site, Saint-etienne-vallee-franc
  - Research Site, Saint-Euphrône
  - Research Site, Saint-Eusèbe
  - Research Site, Saint-Égrève
  - Research Site, Saint-Éloy-les-Mines
  - Research Site, Saint-Étienne-aux-Clos
  - Research Site, Saint-Étienne-à-Arnes
  - Research Site, Saint-Étienne-de-Baïgorry
  - Research Site, Saint-Étienne-de-Mer-Morte
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-du-Bois
  - Research Site, Saint-Étienne-du-Rouvray
  - Research Site, Saint-Étienne-la-Geneste
  - Research Site, Saint-Fargeau-Ponthierry
  - Research Site, Saint-Ferme
  - Research Site, Saint-Féliu-d'Amont
  - Research Site, Saint-Félix-de-Sorgues
  - Research Site, Saint-Florent-le-Vieil
  - Research Site, Saint-Florent-sur-Auzonnet
  - Research Site, Saint-Florentin
  - Research Site, Saint-Floris
  - Research Site, Saint-Fort
  - Research Site, Saint-Front
  - Research Site, Saint-Froult
  - Research Site, Saint-Fulgent
  - Research Site, Saint-Galmier
  - Research Site, Saint-Gatien-des-Bois
  - Research Site, Saint-Genest-Lerpt
  - Research Site, Saint-Gengoux-le-National
  - Research Site, Saint-Geniès-de-Malgoirès
  - Research Site, Saint-Genis-d'Hiersac
  - Research Site, Saint-Genis-Laval
  - Research Site, Saint-Georges
  - Research Site, Saint-Georges-d'Espéranche
  - Research Site, Saint-Georges-de-Didonne
  - Research Site, Saint-Georges-de-Mons
  - Research Site, Saint-Georges-de-Montaigu
  - Research Site, Saint-Georges-de-Reneins
  - Research Site, Saint-Georges-des-Coteaux
  - Research Site, Saint-georges-des-groseill
  - Research Site, Saint-Georges-dOrques
  - Research Site, Saint-Georges-du-Rosay
  - Research Site, Saint-Georges-sur-Baulche
  - Research Site, Saint-Georges-sur-Cher
  - Research Site, Saint-germain-de-marencenn
  - Research Site, Saint-Germain-des-Bois
  - Research Site, Saint-Germain-des-Fossés
  - Research Site, Saint-Germain-du-Corbéis
  - Research Site, Saint-Germain-du-Puy
  - Research Site, Saint-Germain-du-Teil
  - Research Site, Saint-Germain-en-Coglès
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-germain-la-blanche-h
  - Research Site, Saint-Germain-le-Fouilloux
  - Research Site, Saint-Germain-Lembron
  - Research Site, Saint-Germain-les-Belles
  - Research Site, Saint-Germain-sur-Meuse
  - Research Site, Saint-Germain-sur-Morin
  - Research Site, Saint-Germain-Village
  - Research Site, Saint-Gervais-les-Bains
  - Research Site, Saint-Gervasy
  - Research Site, Saint-Gély-du-Fesc
  - Research Site, Saint-Géréon
  - Research Site, Saint-Géry
  - Research Site, Saint-Gilles
  - Research Site, Saint-Gilles-Croix-de-Vie
  - Research Site, Saint-Gilles-Pligeaux
  - Research Site, Saint-Girons
  - Research Site, Saint-Herblain
  - Research Site, Saint-Héand
  - Research Site, Saint-Hilaire
  - Research Site, Saint-Hilaire-Cottes
  - Research Site, Saint-Hilaire-de-Brens
  - Research Site, Saint-Hilaire-de-Riez
  - Research Site, Saint-Hippolyte-de-Caton
  - Research Site, Saint-Jean-Bonnefonds
  - Research Site, Saint-Jean-Cap-Ferrat
  - Research Site, Saint-Jean-d'Angély
  - Research Site, Saint-Jean-d'Angle
  - Research Site, Saint-Jean-d'Estissac
  - Research Site, Saint-Jean-de-Bournay
  - Research Site, Saint-Jean-de-Braye
  - Research Site, Saint-Jean-de-Daye
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-de-Linières
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Jean-de-Monts
  - Research Site, Saint-Jean-de-Sixt
  - Research Site, Saint-Jean-de-Thouars
  - Research Site, Saint-Jean-de-Verges
  - Research Site, Saint-Jean-du-Pin
  - Research Site, Saint-Jean-le-Blanc
  - Research Site, Saint-Jeanvrin
  - Research Site, Saint-Jorioz
  - Research Site, Saint-Julien-du-Sault
  - Research Site, Saint-julien-en-saint-alba
  - Research Site, Saint-Julien-les-Villas
  - Research Site, Saint-julien-sous-les-cote
  - Research Site, Saint-Julien-sur-Reyssouze
  - Research Site, Saint-Junien
  - Research Site, Saint-Just
  - Research Site, Saint-Just-la-Pendue
  - Research Site, Saint-Just-le-Martel
  - Research Site, Saint-Just-Saint-Rambert
  - Research Site, Saint-Langis-lès-Mortagne
  - Research Site, Saint-Lary
  - Research Site, Saint-Laurent
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Laurent-de-la-Prée
  - Research Site, Saint-laurent-de-la-salanq
  - Research Site, Saint-Laurent-de-Mure
  - Research Site, Saint-Laurent-du-Pape
  - Research Site, Saint-Laurent-du-Pont
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Laurent-en-Grandvaux
  - Research Site, Saint-Leu-la-Forêt
  - Research Site, Saint-Léger-sous-Cholet
  - Research Site, Saint-Léger-sur-Dheune
  - Research Site, Saint-Léon-sur-l'Isle
  - Research Site, Saint-Léonard
  - Research Site, Saint-Léonard-de-Noblat
  - Research Site, Saint-Lizier
  - Research Site, Saint-Loubès
  - Research Site, Saint-Loup
  - Research Site, Saint-Loup-Cammas
  - Research Site, Saint-Loup-d'Ordon
  - Research Site, Saint-Lyphard
  - Research Site, Saint-Lys
  - Research Site, Saint-Macoux
  - Research Site, Saint-Magne-de-Castillon
  - Research Site, Saint-Maime
  - Research Site, Saint-Mandé
  - Research Site, Saint-Marc-Jaumegarde
  - Research Site, Saint-Marcel-dArdèche
  - Research Site, Saint-Marcel-lès-Valence
  - Research Site, Saint-Mars-d'Égrenne
  - Research Site, Saint-Mars-d'Outillé
  - Research Site, Saint-Mars-sur-la-Futaie
  - Research Site, Saint-Martial-le-Mont
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-d'Ablois
  - Research Site, Saint-Martin-d'Auxigny
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Martin-de-Bienfaite
  - Research Site, Saint-martin-de-boschervil
  - Research Site, Saint-Martin-de-Crau
  - Research Site, Saint-martin-de-saint-maix
  - Research Site, Saint-Martin-de-Seignanx
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-des-Monts
  - Research Site, Saint-Martin-du-Bois
  - Research Site, Saint-Martin-du-Tertre
  - Research Site, Saint-Martin-la-Méanne
  - Research Site, Saint-Martin-Laguépie
  - Research Site, Saint-Martin-le-Beau
  - Research Site, Saint-Martin-le-Châtel
  - Research Site, Saint-Martin-sur-Lavezon
  - Research Site, Saint-Martin-Vésubie
  - Research Site, Saint-Maur
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice
  - Research Site, Saint-Maurice-de-Gourdans
  - Research Site, Saint-Maurice-de-Lignon
  - Research Site, Saint-Maurice-des-Noues
  - Research Site, Saint-Maurice-Montcouronne
  - Research Site, Saint-maurice-sur-dargoire
  - Research Site, Saint-Max
  - Research Site, Saint-Memmie
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Michel
  - Research Site, Saint-Michel-Chef-Chef
  - Research Site, Saint-michel-l'observatoir
  - Research Site, Saint-Michel-sur-Orge
  - Research Site, Saint-Mihiel
  - Research Site, Saint-Mitre-les-Remparts
  - Research Site, Saint-Montan
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Nazaire-d'Aude
  - Research Site, Saint-Nicolas-aux-Bois
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Nicolas-du-Pélem
  - Research Site, Saint-Nom-la-Bretêche
  - Research Site, Saint-Omer
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Ouen
  - Research Site, Saint-Ouen-l'Aumône
  - Research Site, Saint-Ouen-Marchefroy
  - Research Site, Saint-Paër
  - Research Site, Saint-Pair-sur-Mer
  - Research Site, Saint-Pal-de-Chalencon
  - Research Site, Saint-Pantaléon-de-Larche
  - Research Site, Saint-Pardoux-le-Vieux
  - Research Site, Saint-Pargoire
  - Research Site, Saint-Parize-le-Châtel
  - Research Site, Saint-Parres-aux-Tertres
  - Research Site, Saint-Paterne-Racan
  - Research Site, Saint-Patrice-de-Claids
  - Research Site, Saint-Paul-de-Jarrat
  - Research Site, Saint-Paul-des-Landes
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Paul-Trois-Châteaux
  - Research Site, Saint-Père-en-Retz
  - Research Site, Saint-Pé-de-Bigorre
  - Research Site, Saint-Pée-sur-Nivelle
  - Research Site, Saint-Péravy-la-Colombe
  - Research Site, Saint-Péray
  - Research Site, Saint-Philbert-de-Bouaine
  - Research Site, Saint-Philbert-sur-Orne
  - Research Site, Saint-Piat
  - Research Site, Saint-Pierre-d'Entremont
  - Research Site, Saint-Pierre-d'Oléron
  - Research Site, Saint-Pierre-de-Chignac
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-des-Fleurs
  - Research Site, Saint-Pierre-du-Chemin
  - Research Site, Saint-Pierre-du-Mont
  - Research Site, Saint-Pierre-du-Perray
  - Research Site, Saint-Pierre-la-Cour
  - Research Site, Saint-Pierre-Langers
  - Research Site, Saint-Pierre-lès-Elbeuf
  - Research Site, Saint-Pierre-lès-Nemours
  - Research Site, Saint-Planchers
  - Research Site, Saint-Pol-sur-Mer
  - Research Site, Saint-Pol-sur-Ternoise
  - Research Site, Saint-Poncy
  - Research Site, Saint-Porquier
  - Research Site, Saint-Pourçain-sur-Sioule
  - Research Site, Saint-Pôtan
  - Research Site, Saint-Priest
  - Research Site, Saint-Privat-des-Vieux
  - Research Site, Saint-Privé
  - Research Site, Saint-Prix
  - Research Site, Saint-projet-saint-constan
  - Research Site, Saint-Pryvé-Saint-Mesmin
  - Research Site, Saint-Quentin
  - Research Site, Saint-Quentin-en-Mauges
  - Research Site, Saint-Quentin-Fallavier
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Renan
  - Research Site, Saint-Rémy-de-Sillé
  - Research Site, Saint-Rémy-en-Rollat
  - Research Site, Saint-Rémy-lès-Chevreuse
  - Research Site, Saint-Romain
  - Research Site, Saint-Romain-de-Colbosc
  - Research Site, Saint-Rome-de-Dolan
  - Research Site, Saint-Samson-sur-Rance
  - Research Site, Saint-Saturnin
  - Research Site, Saint-Saturnin-sur-Loire
  - Research Site, Saint-Saulve
  - Research Site, Saint-Sauveur
  - Research Site, Saint-Sauveur-des-Landes
  - Research Site, Saint-Sauveur-sur-Tinée
  - Research Site, Saint-Savinien
  - Research Site, Saint-Sernin
  - Research Site, Saint-Sernin-du-Plain
  - Research Site, Saint-Sever
  - Research Site, Saint-Sever-Calvados
  - Research Site, Saint-Sébastien-de-Morsent
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Sigismond
  - Research Site, Saint-Sorlin-en-Valloire
  - Research Site, Saint-Sulpice
  - Research Site, Saint-Sulpice-de-Royan
  - Research Site, Saint-Sulpice-sur-Risle
  - Research Site, Saint-Sylvain-d'Anjou
  - Research Site, Saint-Symphorien
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saint-Thomas-de-Conac
  - Research Site, Saint-Thurial
  - Research Site, Saint-Thuriau
  - Research Site, Saint-Trojan-les-Bains
  - Research Site, Saint-Urcisse
  - Research Site, Saint-Valery-en-Caux
  - Research Site, Saint-Valery-sur-Somme
  - Research Site, Saint-Valérien
  - Research Site, Saint-Vallier
  - Research Site, Saint-Vallier-de-Thiey
  - Research Site, Saint-Venant
  - Research Site, Saint-Viance
  - Research Site, Saint-Vincent de Paul
  - Research Site, Saint-Vincent-de-Cosse
  - Research Site, Saint-Vincent-de-Tyrosse
  - Research Site, Saint-Vincent-Jalmoutiers
  - Research Site, Saint-Vincent-Rive-d'Olt
  - Research Site, Saint-Wandrille-Rançon
  - Research Site, Saint-Yan
  - Research Site, Saint-Yrieix-sur-Charente
  - Research Site, Saint-Yvoine
  - Research Site, Sainte-Adresse
  - Research Site, Sainte-Bazeille
  - Research Site, Sainte-Christine
  - Research Site, Sainte-Croix-sur-Orne
  - Research Site, Sainte-Croix-Volvestre
  - Research Site, Sainte-Feyre
  - Research Site, Sainte-Foy-lès-Lyon
  - Research Site, Sainte-gauburge-sainte-col
  - Research Site, Sainte-genevieve-sur-argen
  - Research Site, Sainte-Geneviève-des-Bois
  - Research Site, Sainte-Livrade-sur-Lot
  - Research Site, Sainte-Marguerite
  - Research Site, Sainte-Maure-de-Touraine
  - Research Site, Sainte-Maxime
  - Research Site, Sainte-Nathalène
  - Research Site, Sainte-Savine
  - Research Site, Sainte-Scolasse-sur-Sarthe
  - Research Site, Sainte-Soline
  - Research Site, Sainte-Soulle
  - Research Site, Saintes
  - Research Site, Saints
  - Research Site, Salaise-sur-Sanne
  - Research Site, Salies-de-Béarn
  - Research Site, Saligny-sur-Roudon
  - Research Site, Salins-les-Bains
  - Research Site, Sallanches
  - Research Site, Salles-d'Aude
  - Research Site, Salomé
  - Research Site, Salon-de-Provence
  - Research Site, Salon-la-Tour
  - Research Site, Salonnes
  - Research Site, Salouël
  - Research Site, Salviac
  - Research Site, Samadet
  - Research Site, San-Nicolao
  - Research Site, Sanary-sur-Mer
  - Research Site, Sancerre
  - Research Site, Sancey-le-Grand
  - Research Site, Sancoins
  - Research Site, Sangatte
  - Research Site, Sannois
  - Research Site, Saramon
  - Research Site, Saran
  - Research Site, Sarbazan
  - Research Site, Sarcelles
  - Research Site, Sarlat-la-Canéda
  - Research Site, Sarrewerden
  - Research Site, Sarrians
  - Research Site, Sartène
  - Research Site, Sartrouville
  - Research Site, Sarzeau
  - Research Site, Sassenage
  - Research Site, Sauchy-Lestrée
  - Research Site, Saugnac-et-Cambran
  - Research Site, Saujon
  - Research Site, Saulcy-sur-Meurthe
  - Research Site, Saulxures-lès-Nancy
  - Research Site, Saumur
  - Research Site, Saunay
  - Research Site, Sausset-les-Pins
  - Research Site, Sautron
  - Research Site, Sauvian
  - Research Site, Sauvigny-le-Bois
  - Research Site, Saverdun
  - Research Site, Savigné-sur-Lathan
  - Research Site, Savigny
  - Research Site, Savigny-en-Sancerre
  - Research Site, Savigny-le-Temple
  - Research Site, Savigny-lès-Beaune
  - Research Site, Savigny-sur-Braye
  - Research Site, Savigny-sur-Orge
  - Research Site, Savines-le-Lac
  - Research Site, Sceaux
  - Research Site, Schiltigheim
  - Research Site, Schwindratzheim
  - Research Site, Scionzier
  - Research Site, Seclin
  - Research Site, Secondigné-sur-Belle
  - Research Site, Sedan
  - Research Site, Seichamps
  - Research Site, Seignosse
  - Research Site, Selles-sur-Cher
  - Research Site, Selommes
  - Research Site, Seloncourt
  - Research Site, Semur-en-Auxois
  - Research Site, Senlis
  - Research Site, Sennecey-le-Grand
  - Research Site, Senones
  - Research Site, Sens
  - Research Site, Sepmes
  - Research Site, Septeuil
  - Research Site, Septfonds
  - Research Site, Sequedin
  - Research Site, Sermaises
  - Research Site, Sermamagny
  - Research Site, Serre-les-Sapins
  - Research Site, Servaville-Salmonville
  - Research Site, Seurre
  - Research Site, Sevrey
  - Research Site, Sevrier
  - Research Site, Seynod
  - Research Site, Seysses
  - Research Site, Seyssinet-Pariset
  - Research Site, Seyssins
  - Research Site, Sète
  - Research Site, Sèvres
  - Research Site, Sèvres-Anxaumont
  - Research Site, Sées
  - Research Site, Séné
  - Research Site, Séreilhac
  - Research Site, Sérigny
  - Research Site, Sézanne
  - Research Site, Sigean
  - Research Site, Signes
  - Research Site, Sillery
  - Research Site, Sillé-le-Guillaume
  - Research Site, Silly-le-Long
  - Research Site, Simandre
  - Research Site, Simandres
  - Research Site, Simard
  - Research Site, Simiane-Collongue
  - Research Site, Sin-le-Noble
  - Research Site, Sion-les-Mines
  - Research Site, Sisteron
  - Research Site, Six-Fours-les-Plages
  - Research Site, Sochaux
  - Research Site, Soing-Cubry-Charentenay
  - Research Site, Soissons
  - Research Site, Soisy-sous-Montmorency
  - Research Site, Soisy-sur-Seine
  - Research Site, Solaize
  - Research Site, Solesmes
  - Research Site, Sommette-Eaucourt
  - Research Site, Sommeval
  - Research Site, Sonnay
  - Research Site, Sorcy-Saint-Martin
  - Research Site, Sore
  - Research Site, Sorgues
  - Research Site, Sornay
  - Research Site, Sospel
  - Research Site, Sottevast
  - Research Site, Souancé-au-Perche
  - Research Site, Soueich
  - Research Site, Souffelweyersheim
  - Research Site, Soufflenheim
  - Research Site, Sougères-en-Puisaye
  - Research Site, Sougé-le-Ganelon
  - Research Site, Souillac
  - Research Site, Soulac-sur-Mer
  - Research Site, Soulitré
  - Research Site, Soullans
  - Research Site, Soulles
  - Research Site, Soumaintrain
  - Research Site, Soustons
  - Research Site, Souvans
  - Research Site, Souvigny-en-Sologne
  - Research Site, Spéracèdes
  - Research Site, St-Malo
  - Research Site, Stains
  - Research Site, Steene
  - Research Site, Strasbourg
  - Research Site, Subligny
  - Research Site, Sucy-en-Brie
  - Research Site, Suèvres
  - Research Site, Sugères
  - Research Site, Suippes
  - Research Site, Suresnes
  - Research Site, Surgères
  - Research Site, Sury-le-Comtal
  - Research Site, Sussat
  - Research Site, Suze-la-Rousse
  - Research Site, Taillades
  - Research Site, Taillecourt
  - Research Site, Talairan
  - Research Site, Talange
  - Research Site, Talant
  - Research Site, Talcy
  - Research Site, Talence
  - Research Site, Tallenay
  - Research Site, Taller
  - Research Site, Taradeau
  - Research Site, Tarare
  - Research Site, Tarascon
  - Research Site, Tarbes
  - Research Site, Tarnès
  - Research Site, Tarnos
  - Research Site, Tassin-la-Demi-Lune
  - Research Site, Tatinghem
  - Research Site, Taulé
  - Research Site, Tauriac
  - Research Site, Taverny
  - Research Site, Tayac
  - Research Site, Teillé
  - Research Site, Templeuve-en-Pévèle
  - Research Site, Tence
  - Research Site, Tergnier
  - Research Site, Termes-d'Armagnac
  - Research Site, Termignon
  - Research Site, Ternay
  - Research Site, Terrasson-Lavilledieu
  - Research Site, Teurthéville-Hague
  - Research Site, Téteghem
  - Research Site, Theillay
  - Research Site, Thénioux
  - Research Site, Thénorgues
  - Research Site, Thiais
  - Research Site, Thiberville
  - Research Site, Thièvres
  - Research Site, Thionville
  - Research Site, Thizy
  - Research Site, Thonon-les-Bains
  - Research Site, Thorens-Glières
  - Research Site, Thorigné-Fouillard
  - Research Site, Thorigné-sur-Dué
  - Research Site, Thouars
  - Research Site, Thourotte
  - Research Site, Thuir
  - Research Site, Thury-en-Valois
  - Research Site, Tignieu
  - Research Site, Tillières
  - Research Site, Tilloy-lez-Cambrai
  - Research Site, Tilloy-lès-Mofflaines
  - Research Site, Tinqueux
  - Research Site, Tizac-de-Lapouyade
  - Research Site, Tocqueville-les-Murs
  - Research Site, Tollevast
  - Research Site, Tomblaine
  - Research Site, Tonnay-Boutonne
  - Research Site, Tonnay-Charente
  - Research Site, Tonneins
  - Research Site, Tonnerre
  - Research Site, Torcenay
  - Research Site, Torcy
  - Research Site, Tortefontaine
  - Research Site, Tosny
  - Research Site, Tosse
  - Research Site, Toucy
  - Research Site, Toudon
  - Research Site, Toufflers
  - Research Site, Toul
  - Research Site, Toulenne
  - Research Site, Toulon
  - Research Site, Toulon-sur-Allier
  - Research Site, Toulouges
  - Research Site, Toulouse
  - Research Site, Touquin
  - Research Site, Tourcoing
  - Research Site, Tourlaville
  - Research Site, Tournai-sur-Dive
  - Research Site, Tournedos-Bois-Hubert
  - Research Site, Tournefeuille
  - Research Site, Tournes
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tournus
  - Research Site, Tourouvre
  - Research Site, Tours
  - Research Site, Tourville-sur-Sienne
  - Research Site, Toussieu
  - Research Site, Tracy-Bocage
  - Research Site, Traînel
  - Research Site, Trans-en-Provence
  - Research Site, Trans-sur-Erdre
  - Research Site, Trappes
  - Research Site, Tremblay-en-France
  - Research Site, Tremblois-lès-Carignan
  - Research Site, Tresses
  - Research Site, Tressin
  - Research Site, Trédrez-Locquémeau
  - Research Site, Trégomeur
  - Research Site, Trégueux
  - Research Site, Tréguier
  - Research Site, Trélazé
  - Research Site, Trélissac
  - Research Site, Trélon
  - Research Site, Tréméloir
  - Research Site, Trépail
  - Research Site, Trévenans
  - Research Site, Trévoux
  - Research Site, Trézelles
  - Research Site, Trie-la-Ville
  - Research Site, Trie-sur-Baïse
  - Research Site, Trignac
  - Research Site, Trizay
  - Research Site, Troisvilles
  - Research Site, Trosly-Breuil
  - Research Site, Troyes
  - Research Site, Truchtersheim
  - Research Site, Trugny
  - Research Site, Turckheim
  - Research Site, Turenne
  - Research Site, Turny
  - Research Site, Uckange
  - Research Site, Ugine
  - Research Site, Unchair
  - Research Site, Ur
  - Research Site, Urcel
  - Research Site, Urville-Nacqueville
  - Research Site, Ury
  - Research Site, Usseau
  - Research Site, Ussel
  - Research Site, Uxegney
  - Research Site, Vabres-l'Abbaye
  - Research Site, Vacognes-Neuilly
  - Research Site, Vagney
  - Research Site, Vaires-sur-Marne
  - Research Site, Vaison-la-Romaine
  - Research Site, Vaivre-et-Montoille
  - Research Site, Val-de-Meuse
  - Research Site, Val-des-Prés
  - Research Site, Valailles
  - Research Site, Valbonne
  - Research Site, Valdoie
  - Research Site, Valence
  - Research Site, Valence-d'Albigeois
  - Research Site, Valenciennes
  - Research Site, Valentigney
  - Research Site, Valenton
  - Research Site, Vallans
  - Research Site, Vallauris
  - Research Site, Valleroy
  - Research Site, Vallet
  - Research Site, Vallières-les-Grandes
  - Research Site, Vallon-en-Sully
  - Research Site, Vallon-Pont-d'Arc
  - Research Site, Valognes
  - Research Site, Valréas
  - Research Site, Valsemé
  - Research Site, Vandrimare
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Vanves
  - Research Site, Varaire
  - Research Site, Vareilles
  - Research Site, Varennes-sur-Allier
  - Research Site, Varennes-Vauzelles
  - Research Site, Varogne
  - Research Site, Vasles
  - Research Site, Vatilieu
  - Research Site, Vaucouleurs
  - Research Site, Vaudry
  - Research Site, Vaujours
  - Research Site, Vauréal
  - Research Site, Vautorte
  - Research Site, Vauvert
  - Research Site, Vaux
  - Research Site, Vaux-le-Pénil
  - Research Site, Vaux-sur-Mer
  - Research Site, Vauxbuin
  - Research Site, Veauchette
  - Research Site, Veauville-lès-Baons
  - Research Site, Vedène
  - Research Site, Velaux
  - Research Site, Vendat
  - Research Site, Vendays-Montalivet
  - Research Site, Vendenheim
  - Research Site, Vendin-le-Vieil
  - Research Site, Vendôme
  - Research Site, Venizy
  - Research Site, Vennans
  - Research Site, Verberie
  - Research Site, Verdes
  - Research Site, Verdun
  - Research Site, Verdun-sur-le-Doubs
  - Research Site, Verfeil
  - Research Site, Verlinghem
  - Research Site, Vernet
  - Research Site, Verneuil-en-Halatte
  - Research Site, Verneuil-sur-Seine
  - Research Site, Verniolle
  - Research Site, Vernou-la-Celle-sur-Seine
  - Research Site, Vernou-sur-Brenne
  - Research Site, Verny
  - Research Site, Verquin
  - Research Site, Verrières
  - Research Site, Verrières-le-Buisson
  - Research Site, Versailles
  - Research Site, Vert
  - Research Site, Vert-Saint-Denis
  - Research Site, Verton
  - Research Site, Vertou
  - Research Site, Vesc
  - Research Site, Vesoul
  - Research Site, Veynes
  - Research Site, Veyre-Monton
  - Research Site, Veyrins-Thuellin
  - Research Site, Vezin-le-Coquet
  - Research Site, Vezins
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Vézeronce-Curtin
  - Research Site, Vézins-de-Lévézou
  - Research Site, Viarmes
  - Research Site, Vic-sur-Aisne
  - Research Site, Vichy
  - Research Site, Vicq
  - Research Site, Vidauban
  - Research Site, Vidouze
  - Research Site, Viefvillers
  - Research Site, Vieillevigne
  - Research Site, Vielmur-sur-Agout
  - Research Site, Vienne
  - Research Site, Vierzon
  - Research Site, Vieu
  - Research Site, Vieux-Ferrette
  - Research Site, Vif
  - Research Site, Vigneulles-les-hattonchate
  - Research Site, Vigneux-sur-Seine
  - Research Site, Vignevieille
  - Research Site, Vignoux-sur-Barangeon
  - Research Site, Villalier
  - Research Site, Villandry
  - Research Site, Villard-Bonnot
  - Research Site, Villard-de-Lans
  - Research Site, Villars-les-Bois
  - Research Site, Villars-les-Dombes
  - Research Site, Villate
  - Research Site, Villaz
  - Research Site, Ville-la-Grand
  - Research Site, Villebarou
  - Research Site, Villebichot
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villebrumier
  - Research Site, Villecresnes
  - Research Site, Villecroze
  - Research Site, Villefontaine
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejésus
  - Research Site, Villejuif
  - Research Site, Villemagne-l'Argentière
  - Research Site, Villemandeur
  - Research Site, Villemolaque
  - Research Site, Villemomble
  - Research Site, Villemoutiers
  - Research Site, Villenauxe-la-Grande
  - Research Site, Villenave-d'Ornon
  - Research Site, Villenave-près-Béarn
  - Research Site, Villeneuve les beziers
  - Research Site, Villeneuve-d'Ascq
  - Research Site, Villeneuve-de-Berg
  - Research Site, Villeneuve-de-la-Raho
  - Research Site, Villeneuve-de-Marsan
  - Research Site, Villeneuve-de-Rivière
  - Research Site, Villeneuve-la-Garenne
  - Research Site, Villeneuve-le-Comte
  - Research Site, Villeneuve-le-Roi
  - Research Site, Villeneuve-les-Bordes
  - Research Site, Villeneuve-lès-Avignon
  - Research Site, Villeneuve-Loubet
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villeneuve-sur-Yonne
  - Research Site, Villeneuve-Tolosane
  - Research Site, Villeparisis
  - Research Site, Villeparois
  - Research Site, Villepinte
  - Research Site, Villepreux
  - Research Site, Villers-Cotterêts
  - Research Site, Villers-le-Lac
  - Research Site, Villers-lès-Nancy
  - Research Site, Villers-Pol
  - Research Site, Villers-Semeuse
  - Research Site, Villers-sous-Prény
  - Research Site, Villers-sur-Mer
  - Research Site, Villersexel
  - Research Site, Villeurbanne
  - Research Site, Villevieille
  - Research Site, Villiers-Adam
  - Research Site, Villiers-en-Lieu
  - Research Site, Villiers-le-Bel
  - Research Site, Villiers-Saint-Denis
  - Research Site, Villiers-sous-Grez
  - Research Site, Villiers-sur-Marne
  - Research Site, Vinassan
  - Research Site, Vincennes
  - Research Site, Vincey
  - Research Site, Vineuil
  - Research Site, Vinon-sur-Verdon
  - Research Site, Violès
  - Research Site, Viroflay
  - Research Site, Viry
  - Research Site, Viry-Châtillon
  - Research Site, Viry-Noureuil
  - Research Site, Vitrac-sur-Montane
  - Research Site, Vitrey-sur-Mance
  - Research Site, Vitré
  - Research Site, Vitrolles
  - Research Site, Vitry-sur-Orne
  - Research Site, Vitry-sur-Seine
  - Research Site, Vivier-au-Court
  - Research Site, Viviers-du-Lac
  - Research Site, Vivy
  - Research Site, Voiron
  - Research Site, Vollore-Ville
  - Research Site, Volvic
  - Research Site, Voreppe
  - Research Site, Vouillé
  - Research Site, Voujeaucourt
  - Research Site, Vouneuil-sous-Biard
  - Research Site, Vouvray-sur-Loir
  - Research Site, Vouxey
  - Research Site, Vouziers
  - Research Site, Voves
  - Research Site, Vrigne-aux-Bois
  - Research Site, Vuillafans
  - Research Site, Vy-lès-Lure
  - Research Site, Wambrechies
  - Research Site, Wamin
  - Research Site, Warloy-Baillon
  - Research Site, Warmeriville
  - Research Site, Wasquehal
  - Research Site, Wasserbourg
  - Research Site, Watten
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Wemaers-Cappel
  - Research Site, Wignehies
  - Research Site, Wimereux
  - Research Site, Wimille
  - Research Site, Wintzenheim
  - Research Site, Witry-lès-Reims
  - Research Site, Wittelsheim
  - Research Site, Wittenheim
  - Research Site, Wormhout
  - Research Site, Woustviller
  - Research Site, Wulverdinghe
  - Research Site, Xertigny
  - Research Site, Xeuilley
  - Research Site, Xonrupt-Longemer
  - Research Site, Yerres
  - Research Site, Ymeray
  - Research Site, Yssingeaux
  - Research Site, Ytres
  - Research Site, Yutz
  - Research Site, Yves
  - Research Site, Yvetot
  - Research Site, Yville-sur-Seine
  - Research Site, Yvré-l'Évêque
  - Research Site, Yzernay
  - Research Site, Yzeure